CLINICAL TRIAL: NCT02310763
Title: A PHASE 2 RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, MULTIPLE ASCENDING DOSE STUDY TO EVALUATE THE SAFETY, EFFICACY, PHARMACOKINETICS AND PHARMACODYNAMICS OF PF-06252616 IN AMBULATORY BOYS WITH DUCHENNE MUSCULAR DYSTROPHY
Brief Title: A Phase 2 Study to Evaluate the Safety, Efficacy, Pharmacokinetics and Pharmacodynamics of PF-06252616 in Duchenne Muscular Dystrophy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Termination Date 30AUG2018: Reason for termination: Lack of Efficacy
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B5161002; 2014-002072-92 (EudraCT Number)
Record Dates: First submitted 2014-11-04; First posted 2014-12-08 (Estimated); Results first posted 2019-07-23 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-10

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy, myostatin
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — domagrozumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PF-06252616 (Experimental): 3 dose levels (5mg/kg, 20mg/kg and 40 mg/kg) of IV infused PF-06252616 will be investigated within each subject
  Interventions: Biological: PF-06252616
- Placebo (Placebo Comparator): Matching Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: PF-06252616 — PF-06252616 IV Infusion, 3 dose levels (5mg/kg, 20 mg/kg and 40 mg/kg) will be investigated within each subject
  Arms: PF-06252616
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a Phase 2 randomized, 2-period, double-blind, placebo-controlled, multiple ascending dose study to evaluate the safety, efficacy, PK and PD of PF-06252616 administered to ambulatory boys diagnosed with Duchenne Muscular Dystrophy. Three intravenous (IV) dose levels will be investigated in a within subject dose escalating fashion. Subjects will be randomly assigned to 1 of 3 sequence groups for approximately 96 weeks (2 periods of 48 weeks each). In period 1, two of the sequence groups will receive PF-06252616 and one sequence group will receive placebo. In period 2, the placebo group will switch to PF-06252616 and the two remaining sequence groups will either receive placebo or PF-06252616. Efficacy will be based on an observed mean change from baseline on function (4 stair climb) of PF-06252616 as compared to the placebo at the end of period 1. Period 2 provides an opportunity to evaluate PK. Subjects will receive monthly IV infused doses of either PF-06252616 or placebo and will undergo safety evaluations (Laboratory, cardiac monitoring, physical exams, x-ray, MRI), functional evaluations (pulmonary function testing, 4 stair climb, range of motion, strength testing, Northstar Ambulatory Assessment, upper limb functional testing and the six minute walk test), pharmacokinetic testing and pharmacodynamic testing to evaluate changes in muscle volume (MRI).

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory boys age 6 to <16 years old (at the time of randomization), diagnosed with DMD. Diagnosis must be confirmed in subject's medical history and by genetic testing obtained during routine clinical care for diagnostic purposes as reported from an appropriate regulated laboratory using a clinically validated genetic test (genetic testing is not provided by the sponsor).
2. Subjects who are able to perform the 4 stair climb in > or = 0.33 but < or =1.6 stairs/second.
3. Subjects must be receiving glucocorticosteroids for a minimum of 6 months prior to signing informed consent. There should be no significant change (>0.2 mg/kg) in dosage or dose regimen (not related to body weight change) for at least 3 months immediately prior to signing the informed consent and a reasonable expectation that dosage and dosing regimen will not change significantly for the duration of the study.
4. Adequate hepatic and renal function on screening laboratory assessments.
5. No underlying disposition for iron accumulation on screening laboratory assessments.
6. Iron content estimate on the screening liver MRI is within the normal range.

Exclusion Criteria:

1. Subjects with known cognitive impairment or behavioral issues that would impede the ability to follow instructions.
2. History of major surgical procedure within 6 weeks of signing the informed consent or planned surgery during the study.
3. Any injury which may impact functional testing. Previous injuries must be fully healed prior to consenting. Prior lower limb fractures must be fully healed and at least 3 months from injury date.
4. Presence or history of other musculoskeletal or neurologic disease or somatic disorder not related to DMD including pulmonary and cardiac disease.
5. Compromised cardiac function (left ventricular ejection fraction <55% as determined on a screening cardiac MRI or echocardiogram). Subjects may be receiving ACE (angiotensin converting enzyme) inhibitors or beta blockers, ARB (angiotensin II receptor antagonist) or aldosterone blocker/thiazide diuretic; however they must have initiated treatment more than 3 months prior to screening to ensure stable therapy.
6. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular (including uncontrolled hypertension), hepatic, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
7. Documented history of iron overload including hemochromatosis, beta thalassemia major, beta thalassemia intermedia or hemolytic anemia.
8. Unwilling or unable (eg, metal implants, requires sedation) to undergo examination with closed MRI without sedation.
9. Participation in other studies involving investigational drug(s) for a minimum of 30 days or within 5 half lives (whichever is longer) prior to signing the informed consent and/or during study participation.
10. Current or prior treatment with anti-myostatin, exon skipping, nonsense mutation targeted therapies ever or more than 30 days of treatment with utrophin modifiers and treatment with utrophin modifiers within 30 days prior ot signing the informed consent and/or during study participation.
11. Current or prior treatment within the past 3 months with androgens or human growth hormone.
12. Current treatment with immunosuppressant therapies (other than glucocorticoid steroids), aminoglycosides (eg, gentamicin), multi vitamins with iron and iron supplements and other investigational therapies (including idebenone).

Ages: 6 Years to 15 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 121 (Actual)
Dates: Start 2014-11-24 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (65):
- United States (30):
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Ronald Reagan UCLA Pharmacy, Los Angeles, California
  - UCLA (David Geffen School of Medicine), Los Angeles, California
  - University of California, Davis Medical Center, Sacramento, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Shriners Hospitals for Children - Tampa, Tampa, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Iowa ICTS, Iowa City, Iowa
  - KU Clinical Research Center, Clinical and Translational Science Unit(CTSU), Fairway, Kansas
  - University of Kansas-Clinical Research Center, Investigational Pharmacy, Fairway, Kansas
  - University of Kansas Medical Center, Landon Center on Aging, Kansas City, Kansas
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kennedy Krieger Institute Out-patient center, Baltimore, Maryland
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Johns Hopkins Investigational Drug Service, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota Masonic Children's Hospital, Minneapolis, Minnesota
  - St Louis Children's Hospital, St Louis, Missouri
  - Duke University Medical Center,Lenox Baker Children's Hospital, Durham, North Carolina
  - Duke University, Investigational Drug Pharmacy, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Center for Clinical and Translational Sciences, Salt Lake City, Utah
  - Utah Center for Advanced Imaging and Research (UCAIR), Salt Lake City, Utah
  - Investigational Drug Services, Salt Lake City, Utah
  - University of Utah, Department of Neurology, Salt Lake City, Utah
  - University of Utah Medical Center, Salt Lake City, Utah
  - University of Utah School of Medicine, Salt Lake City, Utah
- Lady Cilento Children's Hospital, South Brisbane, Queensland, Australia
- Bulgaria (5):
  - Clinical Densitometry and Bone Metabolic Disease Department, General and Clinical Pathology Clinic, Sofia
  - Hospital Pharmacy, UMHAT Alexandrovska, Sofia
  - Imaging Diagnostic Clinic,UMHAT Alexandrovska, Sofia
  - Neurology Disease Clinic,UMHAT Alexandrovska, Sofia
  - UMHAT Alexandrovska Cardiology Department,Internal Diseases Propaedeutic Clinic, Sofia
- Canada (4):
  - Alberta Children's Hospital, Calgary, Alberta
  - UBC Children's and Women's Health Center of British Columbia, Vancouver, British Columbia
  - Children's Hospital- London Health Sciences Centre, London, Ontario
  - CHU Sainte-Justine, Montreal, Quebec
- Italy (11):
  - UOC Farmacia-Istituto Gianna Gaslini, Istituto Pediatrico di Ricovero e Cura a Carattere Scientifico, Genova
  - UOC Medicina Fisica Riabilitativa, Genova
  - UOC Neurologia Pediatrica e Malattie Muscolari, Genova
  - UOC Radiologia-Istituto Gianna. Gaslini, Istituto Pediatrico di Ricovero e Cura a Carattere, Genova
  - UOS Dipartimentale Endocrinologia Clinica Sperimentale, Genova
  - Dipartimento Pediatrico Universitario-Ospedaliero Endocrinologia, Rome
  - Farmacia Ospedaliera, IRCCS Ospedale Pediatrico Bambino Gesù, Padiglione Sant'Onofrio, Rome
  - Malattie Neuromuscolari e Neurodegenerative, IRCCS Ospedale Pediatrico Bambino Gesù, Rome
  - Ospedale Pediatrico Bambino Gesù - Centro Trial, DPUO - Padiglione Salviati, Rome
  - U.O.C Farmacia, Rome
  - U.O.C. Neuropsichiatria Infantile, Fondazione Policlinico, Rome
- Japan (2):
  - Hyogo college of medicine hospital, Hyōgo
  - National Center of Neurology and Psychiatry, Tokyo
- Poland (6):
  - Samodzielny Publiczny Centralny Szpital Kliniczny w Warszawie Apteka Szpitalna Blok F, Warsaw
  - Samodzielny Publiczny Centralny Szpital Kliniczny w Warszawie, I Katedra i Klinika Kardiologii, Warsaw
  - Samodzielny Publiczny Centralny Szpital Kliniczny w Warszawie, II Zaklad Radiologii Klinicznej, Warsaw
  - Samodzielny Publiczny Centralny Szpital Kliniczny w Warszawie, Klinika Neurologii, Warsaw
  - Samodzielny Publiczny Centralny Szpital Kliniczny w Warszawie, Laboratorium Centralne, Warsaw
  - MTZ Clinical Research Sp.z o.o., Warsaw
- United Kingdom (6):
  - Alder Hey Children's NHS Foundation Trust, Liverpool
  - Dubowitz Neuromuscular Centre Institute of Child Health, London
  - Great Ormond Street Hospital, London
  - Institute of Genetic Medicine, Muscle Team, Newcastle upon Tyne
  - Clinical Research Facility, Newcastle upon Tyne
  - Royal Victoria Infirmary Research Pharmacy, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Sherlock SP, McCrady A, Palmer J, Aghamolaey H, Ahlgren A, Widholm P, Dahlqvist Leinhard O, Karlsson M. Relationship Between Quantitative Magnetic Resonance Imaging Measures and Functional Changes in Patients With Duchenne Muscular Dystrophy. Muscle Nerve. 2025 Mar;71(3):343-352. doi: 10.1002/mus.28321. Epub 2024 Dec 23. PMID 39713935
- [Derived] Sherlock SP, Palmer J, Wagner KR, Abdel-Hamid HZ, Tian C, Mah JK, Muntoni F, Guglieri M, Butterfield RJ, Charnas L, Marraffino S. Dual-energy X-ray absorptiometry measures of lean body mass as a biomarker for progression in boys with Duchenne muscular dystrophy. Sci Rep. 2022 Nov 5;12(1):18762. doi: 10.1038/s41598-022-23072-5. PMID 36335191
- [Derived] Wojciechowski J, Purohit VS, Harnisch LO, Dua P, Tan B, Nicholas T. Population PK and PD Analysis of Domagrozumab in Pediatric Patients with Duchenne Muscular Dystrophy. Clin Pharmacol Ther. 2022 Dec;112(6):1291-1302. doi: 10.1002/cpt.2747. Epub 2022 Oct 4. PMID 36104012
- [Derived] Muntoni F, Guglieri M, Mah JK, Wagner KR, Brandsema JF, Butterfield RJ, McDonald CM, Mayhew AG, Palmer JP, Marraffino S, Charnas L, Mercuri E. Novel approaches to analysis of the North Star Ambulatory Assessment (NSAA) in Duchenne muscular dystrophy (DMD): Observations from a phase 2 trial. PLoS One. 2022 Aug 23;17(8):e0272858. doi: 10.1371/journal.pone.0272858. eCollection 2022. PMID 35998119
- [Derived] Sherlock SP, Palmer J, Wagner KR, Abdel-Hamid HZ, Bertini E, Tian C, Mah JK, Kostera-Pruszczyk A, Muntoni F, Guglieri M, Brandsema JF, Mercuri E, Butterfield RJ, McDonald CM, Charnas L, Marraffino S. Quantitative magnetic resonance imaging measures as biomarkers of disease progression in boys with Duchenne muscular dystrophy: a phase 2 trial of domagrozumab. J Neurol. 2022 Aug;269(8):4421-4435. doi: 10.1007/s00415-022-11084-0. Epub 2022 Apr 8. PMID 35396602
- [Derived] Wagner KR, Guglieri M, Ramaiah SK, Charnas L, Marraffino S, Binks M, Vaidya VS, Palmer J, Goldstein R, Muntoni F. Safety and disease monitoring biomarkers in Duchenne muscular dystrophy: results from a Phase II trial. Biomark Med. 2021 Oct;15(15):1389-1396. doi: 10.2217/bmm-2021-0222. Epub 2021 Sep 17. PMID 34533053
- [Derived] Sherlock SP, Zhang Y, Binks M, Marraffino S. Quantitative muscle MRI biomarkers in Duchenne muscular dystrophy: cross-sectional correlations with age and functional tests. Biomark Med. 2021 Jun;15(10):761-773. doi: 10.2217/bmm-2020-0801. Epub 2021 Jun 22. PMID 34155911
- [Derived] Wagner KR, Abdel-Hamid HZ, Mah JK, Campbell C, Guglieri M, Muntoni F, Takeshima Y, McDonald CM, Kostera-Pruszczyk A, Karachunski P, Butterfield RJ, Mercuri E, Fiorillo C, Bertini ES, Tian C, Statland J, Sadosky AB, Purohit VS, Sherlock SP, Palmer JP, Binks M, Charnas L, Marraffino S, Wong BL. Randomized phase 2 trial and open-label extension of domagrozumab in Duchenne muscular dystrophy. Neuromuscul Disord. 2020 Jun;30(6):492-502. doi: 10.1016/j.nmd.2020.05.002. Epub 2020 May 19. PMID 32522498
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B5161002&StudyName=A%20Phase%202%20Randomized%2C%20Double-blind%2C%20Placebo-controlled%2C%20Multiple%20Ascending%20Dose%20Study%20To%20Evaluate%20The%20Safety%2C%20Efficacy%2C%20Pharmacokinetics%20And%20Pharmacodynamics%20Of%20Pf-06252616%20In%20Ambulatory%20Boys%20With%20Duchenne%20Muscular%20Dystrophy

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 162 participants were screened, 121 participants were enrolled in the study and assigned to 1 of 3 sequences. Only 120 participants received the study treatment and 1 participant withdrew prior to dosing.
Groups:
- Sequence 1: Participants in this sequence received domagrozumab in a dose escalating fashion (5, 20 and 40 mg/kg) for 48 weeks (Period 1). At each dose level, dosing was administered over 2 hours by intravenous infusion every 4 weeks for a total of 16 weeks (4 doses). From Week 49 (Period 2), participants continued to receive domagrozumab at the maximum tolerated dose (40 mg/kg) every 4 weeks for additional 48 weeks or until early termination of the study.
- Sequence 2: Participants in this sequence received domagrozumab in a dose escalating fashion (5, 20 and 40mg/kg) for 48 weeks (Period 1). At each dose level, dosing was administered over 2 hours by intravenous infusion every 4 weeks for a total of 16 weeks (4 doses). From Week 49 (Period 2), participants received placebo for additional 48 weeks or until early termination of the study.
- Sequence 3: Participants in this sequence received placebo for 48 weeks (Period 1). From Week 49 (Period 2), participants received domagrozumab in a dose escalating fashion (5, 20 and 40 mg/kg) for additional 48 weeks or until early termination of the study. At each dose level, dosing was administered over 2 hours by intravenous infusion every 4 weeks for a total of 16 weeks (4 doses).
Period: Period 1 (Weeks 1 to 48)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3
Started | 41 | 39 | 40
Completed | 38 | 37 | 38
Not Completed | 3 | 2 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 1
Not completed — Unable to comply with study procedures | 0 | 1 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Period: Period 2 (Weeks 49 to 96)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3
Started | 38 | 37 | 38
Completed | 22 | 21 | 22
Not Completed | 16 | 16 | 16
Not completed — Study terminated by sponsor | 16 | 16 | 16

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants who received at least 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 41 | 39 | 40 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 41 | 39 | 40 | 120
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.3 (1.9) | 8.5 (1.5) | 9.3 (2.3) | 8.7 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 41 | 39 | 40 | 120
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 33 | 33 | 35 | 101
  Black | 1 | 0 | 1 | 2
  Asian | 6 | 5 | 4 | 15
  Other | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) by Week 49
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a product; the event did not need to have a causal relationship with the treatment. A serious adverse event (SAE) was any untoward medical occurrence at any dose that resulted in death; was life threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in congenital anomaly/birth defect. AEs included both SAEs and AEs. TEAEs were AEs occurred following the start of treatment or AEs increasing in severity during treatment. Severe TEAEs were TEAEs that interfered significantly with participants' usual function. Treatment-related TEAEs were determined by the investigator.
Time Frame: Study Day 1 to Week 49 visit
Population: The analysis population included all participants who received at least 1 dose of investigational drug. Number of participants analyzed signifies number of participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Participants received placebo from Week 1 to Week 48.
- Domagrozumab 5 mg/kg: Participants received domagrozumab at a dose of 5 mg/kg over 2 hours by intravenous infusion every 4 weeks from Week 1 to Week 16 (4 doses).
- Domagrozumab 20 mg/kg: Participants received domagrozumab at a dose of 20 mg/kg over 2 hours by intravenous infusion every 4 weeks from Week 17 to Week 32 (4 doses).
- Domagrozumab 40 mg/kg: Participants received domagrozumab at a dose of 40 mg/kg over 2 hours by intravenous infusion every 4 weeks from Week 33 to Week 48 (4 doses).
Arm/Group | Placebo | Domagrozumab 5 mg/kg | Domagrozumab 20 mg/kg | Domagrozumab 40 mg/kg
Number analyzed (Participants) | 40 | 80 | 78 | 76
Participants
  All-causalities TEAE | 38 | 66 | 57 | 59
  Treatment-related TEAE | 14 | 18 | 14 | 16
  All-causalities serious TEAE | 0 | 1 | 1 | 1
  Treatment-related serious TEAE | 0 | 0 | 0 | 1
  All-causalities severe TEAE | 2 | 2 | 3 | 2
  Treatment-related severe TEAE | 0 | 0 | 0 | 1

2. Primary Outcome: Number of Participants Who Discontinued From the Study Due to TEAEs by Week 49
Description: An AE was any untoward medical occurrence in a clinical investigation participant administered a product; the event did not need to have a causal relationship with the treatment. TEAEs were AEs occurred following the start of treatment or AEs increasing in severity during treatment. Treatment-related TEAEs were determined by the investigator.
Time Frame: Study Day 1 to Week 49 visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Domagrozumab 5 mg/kg | Domagrozumab 20 mg/kg | Domagrozumab 40 mg/kg
Number analyzed (Participants) | 40 | 80 | 78 | 76
Participants
  All-causalities TEAE | 0 | 0 | 0 | 1
  Treatment-related TEAE | 0 | 0 | 0 | 1

3. Primary Outcome: Number of Participants With Dose Reduced or Temporary Discontinuation Due to TEAEs by Week 49
Description: as for outcome 2
Time Frame: Study Day 1 to Week 49 visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Domagrozumab 5 mg/kg | Domagrozumab 20 mg/kg | Domagrozumab 40 mg/kg
Number analyzed (Participants) | 40 | 80 | 78 | 76
Participants
  All-causalities TEAE | 8 | 4 | 4 | 0
  Treatment-related TEAE | 3 | 0 | 1 | 0

4. Primary Outcome: Number of Participants With Laboratory Test Abnormalities (Without Regard to Baseline Abnormality) by Week 49 - Hematology
Description: Hematology evaluation included: hemoglobin, hematocrit, red blood cell (RBC) count, platelets, RBC morphology, white blood cell (WBC) count, absolute lymphocytes, absolute atypical lymphocytes, absolute total neutrophils, absolute total neutrophils count, absolute band cells, absolute basophils, absolute eosinophils, absolute monocytes and absolute myelocytes.
Time Frame: Baseline to Week 49 visit
Population: This analysis population included all participants who received at least 1 dose of investigational drug. Number of participants analyzed signifies number of participants who were evaluable for this outcome measure. Number analyzed refers to number of participants evaluable for specified rows of categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Domagrozumab 5 mg/kg | Domagrozumab 20 mg/kg | Domagrozumab 40 mg/kg
Number analyzed (Participants) | 40 | 80 | 78 | 76
Participants
  Hemoglobin <0.8*lower limit of normal (LLN) | 0 | 0 | 0 | 0
  Hematocrit <0.8*LLN | 0 | 0 | 0 | 0
  RBC count <0.8*LLN | 0 | 0 | 0 | 0
  Platelets <0.5*LLN | 1 | 1 | 1 | 1
  Platelets >1.75*upper limit of normal (ULN) | 0 | 0 | 0 | 0
  RBC Morphology >0 | 0 | 0 | 1 | 1
  WBC count <0.6*LLN | 0 | 0 | 0 | 0
  WBC count >1.5*ULN | 0 | 1 | 1 | 0
  Absolute Lymphocytes <0.8*LLN | 0 | 2 | 2 | 0
  Absolute lymphocytes >1.2*ULN | 1 | 1 | 0 | 0
  Absolute atypical lymphocytes >0 (10*3/uL): number analyzed (Participants) | 0 | 1 | 0 | 1
  Absolute atypical lymphocytes >0 (10*3/uL) |  | 1 |  | 1
  Absolute total neutrophils <0.8*LLN | 1 | 0 | 0 | 0
  Absolute total neutrophils >1.2*ULN | 13 | 8 | 5 | 5
  Absolute total neutrophils count <1.35 (10*3/uL) | 2 | 0 | 2 | 1
  Absolute total neutrophils count >8.15 (10*3/uL) | 20 | 13 | 12 | 9
  Absolute band cells >0.27 (10*3/uL) | 0 | 0 | 0 | 0
  Absolute basophils >1.2*ULN | 2 | 1 | 1 | 2
  Absolute eosinophils >1.2*ULN | 6 | 2 | 6 | 6
  Absolute monocytes >1.2*ULN | 1 | 1 | 2 | 2
  Absolute myelocytes >0 (10*3/uL): number analyzed (Participants) | 0 | 0 | 0 | 1
  Absolute myelocytes >0 (10*3/uL) |  |  |  | 1

5. Primary Outcome: Number of Participants With Laboratory Test Abnormalities (Without Regard to Baseline Abnormality) by Week 49 - Coagulation
Description: Coagulation evaluation included activated partial thromboplastin time (aPTT) and prothrombin time (PT).
Time Frame: Baseline to Week 49 visit
Population: This analysis population included all participants who received at least 1 dose of investigational drug. Number of participants analyzed signifies number of participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Domagrozumab 5 mg/kg | Domagrozumab 20 mg/kg | Domagrozumab 40 mg/kg
Number analyzed (Participants) | 40 | 80 | 78 | 76
Participants
  aPTT >1.1*ULN | 1 | 1 | 1 | 2
  PT >1.1*ULN | 13 | 6 | 3 | 7

6. Primary Outcome: Number of Participants With Laboratory Test Abnormalities (Without Regard to Baseline Abnormality) by Week 49 - Liver Function
Description: Liver function evaluation included: total/direct/indirect bilirubin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma-glutamyl transferase (GGT), alkaline phosphatase, total protein, albumin and glutamate dehydrogenase.
Time Frame: Baseline to Week 49 visit
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Domagrozumab 5 mg/kg | Domagrozumab 20 mg/kg | Domagrozumab 40 mg/kg
Number analyzed (Participants) | 40 | 80 | 78 | 76
Participants
  Total bilirubin >1.5*ULN | 0 | 0 | 0 | 0
  Direct bilirubin >1.5*ULN: number analyzed (Participants) | 1 | 0 | 0 | 1
  Direct bilirubin >1.5*ULN | 0 |  |  | 0
  Indirect bilirubin >1.5*ULN: number analyzed (Participants) | 1 | 0 | 0 | 1
  Indirect bilirubin >1.5*ULN | 0 |  |  | 0
  AST >3*ULN | 39 | 80 | 76 | 74
  ALT >3*ULN | 40 | 80 | 78 | 75
  GGT >3*ULN | 0 | 0 | 0 | 0
  Alkaline phosphatase >3*ULN | 0 | 0 | 0 | 0
  Total protein <0.8*LLN | 0 | 0 | 0 | 0
  Total protein >1.2*ULN | 0 | 0 | 0 | 0
  Albumin <0.8*LLN | 0 | 0 | 0 | 0
  Albumin >1.2*ULN | 0 | 0 | 0 | 0
  Glutamate dehydrogenase >1.0*ULN | 8 | 8 | 6 | 5

7. Primary Outcome: Number of Participants With Laboratory Test Abnormalities (Without Regard to Baseline Abnormality) by Week 49 - Renal Function
Description: Renal function evaluation included: blood urea nitrogen (BUN), creatinine and uric acid.
Time Frame: Baseline to Week 49 visit
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Domagrozumab 5 mg/kg | Domagrozumab 20 mg/kg | Domagrozumab 40 mg/kg
Number analyzed (Participants) | 40 | 80 | 78 | 76
Participants
  BUN >1.3*ULN | 0 | 0 | 0 | 0
  Creatinine >1.3*ULN | 0 | 0 | 0 | 0
  Uric acid >1.2*ULN | 0 | 1 | 3 | 3

8. Primary Outcome: Number of Participants With Laboratory Test Abnormalities (Without Regard to Baseline Abnormality) by Week 49 - Electrolytes
Description: Electrolytes evaluation included: sodium, potassium, chloride, calcium, phosphate, bicarbonate, ferritin, transferrin saturation, iron, iron binding capacity and unsaturated iron binding capacity. Number of participants with iron abnormalities was reported in different age groups.
Time Frame: Baseline to Week 49 visit
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Domagrozumab 5 mg/kg | Domagrozumab 20 mg/kg | Domagrozumab 40 mg/kg
Number analyzed (Participants) | 40 | 80 | 78 | 76
Participants
  Sodium <0.95*LLN | 0 | 0 | 0 | 0
  Sodium >1.05*ULN | 0 | 0 | 0 | 0
  Potassium <0.9*LLN | 0 | 0 | 0 | 0
  Potassium >1.1*ULN | 0 | 0 | 0 | 0
  Chloride <0.9*LLN | 0 | 0 | 0 | 0
  Chloride >1.1*ULN | 0 | 0 | 0 | 0
  Calcium <0.9*LLN | 0 | 0 | 0 | 0
  Calcium >1.1*ULN | 0 | 0 | 0 | 0
  Phosphate <0.8*LLN | 0 | 0 | 0 | 0
  Phosphate >1.2*ULN | 0 | 0 | 0 | 0
  Bicarbonate <0.9*LLN | 8 | 2 | 3 | 4
  Bicarbonate >1.1*ULN | 1 | 0 | 0 | 0
  Iron (1 Year<=Age<11 Years) <50 (ug/dL): number analyzed (Participants) | 31 | 69 | 68 | 65
  Iron (1 Year<=Age<11 Years) <50 (ug/dL) | 19 | 23 | 14 | 11
  Iron (1 Year<=Age<11 Years) >120 (ug/dL): number analyzed (Participants) | 31 | 69 | 68 | 65
  Iron (1 Year<=Age<11 Years) >120 (ug/dL) | 12 | 29 | 33 | 39
  Iron (11 Years<=Age<18 Years) <50 (ug/dL): number analyzed (Participants) | 11 | 11 | 12 | 11
  Iron (11 Years<=Age<18 Years) <50 (ug/dL) | 2 | 4 | 2 | 2
  Iron (11 Years<=Age<18 Years) >170 (ug/dL): number analyzed (Participants) | 11 | 11 | 12 | 11
  Iron (11 Years<=Age<18 Years) >170 (ug/dL) | 0 | 1 | 1 | 0
  Ferritin <15 (ug/L) | 20 | 32 | 38 | 42
  Ferritin >140 (ug/L) | 1 | 1 | 0 | 0
  Iron binding capacity <37.6 (ug/dL) | 0 | 0 | 0 | 0
  Unsaturated iron binding capacity<130 (ug/dL) | 3 | 7 | 6 | 10
  Unsaturated iron binding capacity >375 (ug/dL) | 1 | 0 | 0 | 0
  Transferrin saturation <20% | 26 | 34 | 26 | 20
  Transferrin saturation >50% | 4 | 9 | 19 | 18

9. Primary Outcome: Number of Participants With Laboratory Test Abnormalities (Without Regard to Baseline Abnormality) by Week 49 - Hormones
Description: Hormone evaluations included free thyroxine (T4), thyroid stimulating hormone (TSH), lutenizing hormone (LH), follicle stimulating hormone (FSH), and androstenedione. Numbers of participants with abnormalities of LH, FSH and androstenedione were reported in different age groups.
Time Frame: Baseline to Week 49 visit
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Domagrozumab 5 mg/kg | Domagrozumab 20 mg/kg | Domagrozumab 40 mg/kg
Number analyzed (Participants) | 40 | 80 | 78 | 76
Participants
  Free T4 <0.8*LLN: number analyzed (Participants) | 40 | 77 | 75 | 72
  Free T4 <0.8*LLN | 0 | 0 | 0 | 0
  Free T4 >1.2*ULN: number analyzed (Participants) | 40 | 77 | 75 | 72
  Free T4 >1.2*ULN | 0 | 0 | 0 | 0
  TSH <0.8*LLN: number analyzed (Participants) | 40 | 78 | 75 | 72
  TSH <0.8*LLN | 0 | 2 | 0 | 1
  TSH >1.2*ULN: number analyzed (Participants) | 40 | 78 | 75 | 72
  TSH >1.2*ULN | 0 | 0 | 0 | 0
  LH (15 Days<=Age<7 Years) <0.3 (mIU/mL): number analyzed (Participants) | 2 | 4 | 2 | 0
  LH (15 Days<=Age<7 Years) <0.3 (mIU/mL) | 1 | 2 | 0 |
  LH (15 Days<=Age<7 Years) >2.8 (mIU/mL): number analyzed (Participants) | 2 | 4 | 2 | 0
  LH (15 Days<=Age<7 Years) >2.8 (mIU/mL) | 0 | 0 | 0 |
  LH (7 Years<=Age<9 Years) <0.3 (mIU/mL): number analyzed (Participants) | 10 | 35 | 29 | 24
  LH (7 Years<=Age<9 Years) <0.3 (mIU/mL) | 6 | 23 | 21 | 14
  LH (7 Years<=Age<9 Years) >2.8 (mIU/mL): number analyzed (Participants) | 10 | 35 | 29 | 24
  LH (7 Years<=Age<9 Years) >2.8 (mIU/mL) | 0 | 0 | 0 | 0
  LH (9 Years<=Age<11 Years) <0.3 (mIU/mL): number analyzed (Participants) | 22 | 27 | 33 | 38
  LH (9 Years<=Age<11 Years) <0.3 (mIU/mL) | 17 | 17 | 23 | 27
  LH (9 Years<=Age<11 Years) >2.8 (mIU/mL): number analyzed (Participants) | 22 | 27 | 33 | 38
  LH (9 Years<=Age<11 Years) >2.8 (mIU/mL) | 0 | 0 | 0 | 0
  LH (11 Years<=Age<12 Years) <0.3 (mIU/mL): number analyzed (Participants) | 3 | 3 | 5 | 3
  LH (11 Years<=Age<12 Years) <0.3 (mIU/mL) | 2 | 2 | 3 | 1
  LH (11 Years<=Age<12 Years) >1.8 (mIU/mL): number analyzed (Participants) | 3 | 3 | 5 | 3
  LH (11 Years<=Age<12 Years) >1.8 (mIU/mL) | 1 | 1 | 0 | 0
  LH (12 Years<=Age<13 Years) <0.3 (mIU/mL): number analyzed (Participants) | 4 | 3 | 3 | 2
  LH (12 Years<=Age<13 Years) <0.3 (mIU/mL) | 1 | 1 | 2 | 2
  LH (12 Years<=Age<13 Years) >4.0 (mIU/mL): number analyzed (Participants) | 4 | 3 | 3 | 2
  LH (12 Years<=Age<13 Years) >4.0 (mIU/mL) | 0 | 0 | 0 | 0
  LH (13 Years<=Age<14 Years) <0.3 (mIU/mL): number analyzed (Participants) | 5 | 4 | 2 | 4
  LH (13 Years<=Age<14 Years) <0.3 (mIU/mL) | 3 | 1 | 0 | 1
  LH (13 Years<=Age<14 Years) >6.0 (mIU/mL): number analyzed (Participants) | 5 | 4 | 2 | 4
  LH (13 Years<=Age<14 Years) >6.0 (mIU/mL) | 0 | 1 | 1 | 1
  FSH (4 Years<=Age<7 Years) >6.70 (mIU/mL): number analyzed (Participants) | 2 | 4 | 2 | 0
  FSH (4 Years<=Age<7 Years) >6.70 (mIU/mL) | 0 | 0 | 0 |
  FSH (7 Years<=Age<9 Years) >4.10 (mIU/mL): number analyzed (Participants) | 10 | 35 | 29 | 24
  FSH (7 Years<=Age<9 Years) >4.10 (mIU/mL) | 0 | 0 | 0 | 0
  FSH (9 Years<=Age<11 Years) >4.50 (mIU/mL): number analyzed (Participants) | 22 | 27 | 33 | 38
  FSH (9 Years<=Age<11 Years) >4.50 (mIU/mL) | 0 | 0 | 0 | 0
  FSH (11 Years<=Age<12 Years) <0.40 (mIU/mL): number analyzed (Participants) | 3 | 3 | 5 | 3
  FSH (11 Years<=Age<12 Years) <0.40 (mIU/mL) | 0 | 0 | 0 | 0
  FSH (11 Years<=Age<12 Years) >8.90 (mIU/mL): number analyzed (Participants) | 3 | 3 | 5 | 3
  FSH (11 Years<=Age<12 Years) >8.90 (mIU/mL) | 0 | 0 | 0 | 0
  FSH (12 Years<=Age<13 Years) <0.50 (mIU/mL): number analyzed (Participants) | 4 | 3 | 3 | 2
  FSH (12 Years<=Age<13 Years) <0.50 (mIU/mL) | 0 | 0 | 0 | 0
  FSH (12 Years<=Age<13 Years) >10.50 (mIU/mL): number analyzed (Participants) | 4 | 3 | 3 | 2
  FSH (12 Years<=Age<13 Years) >10.50 (mIU/mL) | 0 | 0 | 0 | 0
  FSH (13 Years<=Age<14 Years) <0.70 (mIU/mL): number analyzed (Participants) | 5 | 4 | 2 | 4
  FSH (13 Years<=Age<14 Years) <0.70 (mIU/mL) | 0 | 1 | 0 | 2
  FSH (13 Years<=Age<14 Years) >10.80 (mIU/mL): number analyzed (Participants) | 5 | 4 | 2 | 4
  FSH (13 Years<=Age<14 Years) >10.80 (mIU/mL) | 0 | 0 | 0 | 0
  Androstenedione (1 Year<=Age<7 Years) <8 (ng/dL): number analyzed (Participants) | 2 | 5 | 2 | 0
  Androstenedione (1 Year<=Age<7 Years) <8 (ng/dL) | 1 | 2 | 1 |
  Androstenedione (1 Year<=Age<7Years) >50(ng/dL): number analyzed (Participants) | 2 | 5 | 2 | 0
  Androstenedione (1 Year<=Age<7Years) >50(ng/dL) | 0 | 0 | 0 |
  Androstenedione (7 Years<=Age<10Years)<3(ng/dL): number analyzed (Participants) | 20 | 49 | 46 | 44
  Androstenedione (7 Years<=Age<10Years)<3(ng/dL) | 5 | 11 | 10 | 7
  Androstenedione(7Years<=Age<10Years) >31(ng/dL): number analyzed (Participants) | 20 | 49 | 46 | 44
  Androstenedione(7Years<=Age<10Years) >31(ng/dL) | 1 | 0 | 4 | 4
  Androstenedione(10Years<=Age<12Years) <7(ng/dL): number analyzed (Participants) | 20 | 16 | 20 | 23
  Androstenedione(10Years<=Age<12Years) <7(ng/dL) | 13 | 8 | 8 | 10
  Androstenedione (10Years<=Age<12Years)>41 (ng/dL): number analyzed (Participants) | 20 | 16 | 20 | 23
  Androstenedione (10Years<=Age<12Years)>41 (ng/dL) | 3 | 0 | 0 | 0
  Androstenedione (12Years<=Age<14Years)<11 (ng/dL): number analyzed (Participants) | 6 | 7 | 5 | 6
  Androstenedione (12Years<=Age<14Years)<11 (ng/dL) | 3 | 4 | 2 | 2
  Androstenedione(12 Years<=Age<14Years)>64 (ng/dL): number analyzed (Participants) | 6 | 7 | 5 | 6
  Androstenedione(12 Years<=Age<14Years)>64 (ng/dL) | 0 | 0 | 0 | 0

10. Primary Outcome: Number of Participants With Laboratory Test Abnormalities (Without Regard to Baseline Abnormality) by Week 49 - Clinical Chemistry
Description: Clinical chemistry evaluation included glucose, creatine kinase (CK), troponin I, and amylase.
Time Frame: Baseline to Week 49 visit
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Domagrozumab 5 mg/kg | Domagrozumab 20 mg/kg | Domagrozumab 40 mg/kg
Number analyzed (Participants) | 40 | 80 | 78 | 76
Participants
  Glucose <0.6*LLN | 0 | 0 | 0 | 0
  Glucose >1.5*ULN | 0 | 1 | 0 | 2
  CK >2.0*ULN | 40 | 80 | 78 | 76
  Troponin I >3.0*ULN: number analyzed (Participants) | 40 | 79 | 74 | 72
  Troponin I >3.0*ULN | 11 | 12 | 10 | 13
  Amylase >1.5*ULN | 0 | 0 | 0 | 1

11. Primary Outcome: Number of Participants With Laboratory Test Abnormalities (Without Regard to Baseline Abnormality) by Week 49 - Urinalysis
Description: Urinalysis included: urine pH, qualitative urine glucose, qualitative urine ketones, qualitative urine protein, qualitative blood/hemoglobin, urine nitrite, urine leukocytes, urine RBC, urine WBC, urine granular casts, urine hyaline casts, urine urate (uric acid) acidic crystal, urine calcium oxalate crystals, urine amorphous crystals, urine bacteria, urine microscopic exam.
Time Frame: Baseline to Week 49 visit
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Domagrozumab 5 mg/kg | Domagrozumab 20 mg/kg | Domagrozumab 40 mg/kg
Number analyzed (Participants) | 40 | 80 | 78 | 76
Participants
  Qualitative urine glucose (dipstick) >=1 | 1 | 0 | 0 | 0
  Qualitative urine ketones(dipstick) >=1 | 3 | 3 | 5 | 6
  Qualitative urine protein (dipstick) >=1 | 0 | 1 | 0 | 0
  Qualitative urine blood/hemoglobin (dipstick) >=1 | 0 | 2 | 1 | 0
  Urine nitrite (dipstick) >=1 | 0 | 0 | 0 | 0
  Urine leukocytes (dipstick): +1 | 0 | 0 | 1 | 1
  Urine RBC >=20 (/high power field[HPF]): number analyzed (Participants) | 14 | 28 | 30 | 22
  Urine RBC >=20 (/high power field[HPF]) | 0 | 0 | 0 | 0
  Urine WBC >=20 (/HPF): number analyzed (Participants) | 25 | 42 | 43 | 38
  Urine WBC >=20 (/HPF) | 0 | 0 | 0 | 0
  Urine granular casts >1 (/low power field [LPF]): number analyzed (Participants) | 1 | 0 | 0 | 0
  Urine granular casts >1 (/low power field [LPF]) | 1 |  |  |
  Urine hyaline casts >1 (/LPF): number analyzed (Participants) | 2 | 0 | 0 | 0
  Urine hyaline casts >1 (/LPF) | 2 |  |  |
  Urine urate (uric acid) acidic crystal: Present: number analyzed (Participants) | 4 | 2 | 2 | 2
  Urine urate (uric acid) acidic crystal: Present | 4 | 2 | 2 | 2
  Urine calcium oxalate crystals: Present: number analyzed (Participants) | 19 | 24 | 23 | 24
  Urine calcium oxalate crystals: Present | 19 | 24 | 23 | 24
  Urine amorphous crystals: Present: number analyzed (Participants) | 7 | 7 | 6 | 11
  Urine amorphous crystals: Present | 7 | 7 | 6 | 11
  Urine bacteria >20 (/HPF): number analyzed (Participants) | 5 | 4 | 5 | 5
  Urine bacteria >20 (/HPF) | 0 | 0 | 0 | 0
  Urine microscopic exam: Positive: number analyzed (Participants) | 31 | 55 | 52 | 46
  Urine microscopic exam: Positive | 31 | 50 | 49 | 45
  Urine pH (dipstick) <4.5 | 0 | 0 | 0 | 0
  Urine pH (dipstick) >8 | 0 | 1 | 1 | 1

12. Primary Outcome: Number of Participants With Laboratory Test Abnormalities (Without Regard to Baseline Abnormality) by Week 49 - Fecal
Description: Number of participants with blood detected in fecal samples is presented.
Time Frame: Baseline to Week 49 visit
Population: This analysis population included all participants who received at least 1 dose of investigational drug and had at least 1 fecal evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Domagrozumab 5 mg/kg | Domagrozumab 20 mg/kg | Domagrozumab 40 mg/kg
Number analyzed (Participants) | 40 | 79 | 78 | 74
Participants | 2 | 8 | 2 | 3

13. Primary Outcome: Categorical Summary of Liver Iron Accumulation by Week 49
Description: Magnetic resonance imaging (MRI) of Liver was obtained to quantify liver iron accumulation for safety monitoring. MRIs were sent to an independent central radiology imaging facility for calculation of the average transverse relaxation rate (R2*) value which was used to monitor for iron accumulation in the liver. Number of participants meeting the following criteria is presented as follows: 1) normal: R2*<=75Hz at 1.5T or <=139 Hz at 3.0T; 2) above normal: R2*>75Hz and <=190Hz at 1.5T or R2* >139Hz and <=369Hz at 3.0T; 3) mild overload: R2*>190Hz at 1.5T or R2*>360Hz at 3.0T.
Time Frame: Screening, Weeks 13, 29 and 45
Population: This analysis population included all participants who received at least 1 dose of investigational drug. Number analyzed refers to number of participants evaluable for specified rows of categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3
Number analyzed (Participants) | 41 | 39 | 40
Participants
  Normal, Screening | 41 | 39 | 40
  Above normal, Screening | 0 | 0 | 0
  Mild overload, Screening | 0 | 0 | 0
  Normal, Week 13: number analyzed (Participants) | 27 | 24 | 26
  Normal, Week 13 | 27 | 24 | 26
  Above normal, Week 13: number analyzed (Participants) | 27 | 24 | 26
  Above normal, Week 13 | 0 | 0 | 0
  Mild overload, Week 13: number analyzed (Participants) | 27 | 24 | 26
  Mild overload, Week 13 | 0 | 0 | 0
  Normal, Week 29: number analyzed (Participants) | 23 | 21 | 21
  Normal, Week 29 | 23 | 21 | 21
  Above normal, Week 29: number analyzed (Participants) | 23 | 21 | 21
  Above normal, Week 29 | 0 | 0 | 0
  Mild overload, Week 29: number analyzed (Participants) | 23 | 21 | 21
  Mild overload, Week 29 | 0 | 0 | 0
  Normal, Week 45: number analyzed (Participants) | 37 | 37 | 38
  Normal, Week 45 | 37 | 37 | 38
  Above normal, Week 45: number analyzed (Participants) | 37 | 37 | 38
  Above normal, Week 45 | 0 | 0 | 0
  Mild overload, Week 45: number analyzed (Participants) | 37 | 37 | 38
  Mild overload, Week 45 | 0 | 0 | 0

14. Primary Outcome: Number of Participants With Physical Examination Findings Reported as SAEs by Week 49
Description: Physical examination included head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, gastrointestinal, musculoskeletal, and neurological systems. A targeted nose and throat mucosal exam were also performed to monitor for any signs of mucosal telangiectasias. An SAE was any untoward medical occurrence at any dose that resulted in death; was life threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in congenital anomaly/birth defect. Investigators determined which physical examination findings were reported as SAEs.
Time Frame: Baseline to Week 49 visit
Population: This analysis population included all participants who received at least 1 dose of investigational drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3
Number analyzed (Participants) | 41 | 39 | 40
Participants | 0 | 0 | 0

15. Primary Outcome: Summary of Tanner Stage Rating by Week 49
Description: Tanner staging was performed before the first dose of each dose escalation to monitor for signs of accelerated sexual development. The physical changes in pubertal development (pubic hair, penis and testes) were assessed using the system described by Marshall and Tanner. Stage 1 is preadolescent, Stages 2, 3, and 4 are initiation of puberty and Stage 5 is mature adult. Details about the system can be referred to Tanner JM. Growth at Adolescence. Blackwell Scientific Publications 1962; 2nd edition.
Time Frame: Baseline, Weeks 17, 33 and 49
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Groups:
- Domagrozumab: Participants received domagrozumab in a dose escalating fashion (5, 20 and 40mg/kg) from Week 1 to Week 48. At each dose level, dosing was administered over 2 hours by intravenous infusion every 4 weeks for a total of 16 weeks (4 doses).
Arm/Group | Placebo | Domagrozumab
Number analyzed (Participants) | 40 | 80
Participants
  Pubic hair, Stage 1, Baseline: number analyzed (Participants) | 40 | 78
  Pubic hair, Stage 1, Baseline | 35 | 70
  Pubic hair, Stage 2, Baseline: number analyzed (Participants) | 40 | 78
  Pubic hair, Stage 2, Baseline | 4 | 7
  Pubic hair, Stage 3, Baseline: number analyzed (Participants) | 40 | 78
  Pubic hair, Stage 3, Baseline | 0 | 1
  Pubic hair, Stage 4, Baseline: number analyzed (Participants) | 40 | 78
  Pubic hair, Stage 4, Baseline | 1 | 0
  Pubic hair, Stage 5, Baseline: number analyzed (Participants) | 40 | 78
  Pubic hair, Stage 5, Baseline | 0 | 0
  Pubic hair, Stage 1, Week 17: number analyzed (Participants) | 40 | 77
  Pubic hair, Stage 1, Week 17 | 30 | 64
  Pubic hair, Stage 2, Week 17: number analyzed (Participants) | 40 | 77
  Pubic hair, Stage 2, Week 17 | 9 | 11
  Pubic hair, Stage 3, Week 17: number analyzed (Participants) | 40 | 77
  Pubic hair, Stage 3, Week 17 | 0 | 2
  Pubic hair, Stage 4, Week 17: number analyzed (Participants) | 40 | 77
  Pubic hair, Stage 4, Week 17 | 1 | 0
  Pubic hair, Stage 5, Week 17: number analyzed (Participants) | 40 | 77
  Pubic hair, Stage 5, Week 17 | 0 | 0
  Pubic hair, Stage 1, Week 33: number analyzed (Participants) | 36 | 75
  Pubic hair, Stage 1, Week 33 | 23 | 60
  Pubic hair, Stage 2, Week 33: number analyzed (Participants) | 36 | 75
  Pubic hair, Stage 2, Week 33 | 11 | 13
  Pubic hair, Stage 3, Week 33: number analyzed (Participants) | 36 | 75
  Pubic hair, Stage 3, Week 33 | 1 | 1
  Pubic hair, Stage 4, Week 33: number analyzed (Participants) | 36 | 75
  Pubic hair, Stage 4, Week 33 | 1 | 1
  Pubic hair, Stage 5, Week 33: number analyzed (Participants) | 36 | 75
  Pubic hair, Stage 5, Week 33 | 0 | 0
  Pubic hair, Stage 1, Week 49: number analyzed (Participants) | 37 | 72
  Pubic hair, Stage 1, Week 49 | 21 | 52
  Pubic hair, Stage 2, Week 49: number analyzed (Participants) | 37 | 72
  Pubic hair, Stage 2, Week 49 | 11 | 15
  Pubic hair, Stage 3, Week 49: number analyzed (Participants) | 37 | 72
  Pubic hair, Stage 3, Week 49 | 3 | 4
  Pubic hair, Stage 4, Week 49: number analyzed (Participants) | 37 | 72
  Pubic hair, Stage 4, Week 49 | 1 | 1
  Pubic hair, Stage 5, Week 49: number analyzed (Participants) | 37 | 72
  Pubic hair, Stage 5, Week 49 | 1 | 0
  Penis, Stage 1, Baseline: number analyzed (Participants) | 40 | 78
  Penis, Stage 1, Baseline | 30 | 70
  Penis, Stage 2, Baseline: number analyzed (Participants) | 40 | 78
  Penis, Stage 2, Baseline | 9 | 7
  Penis, Stage 3, Baseline: number analyzed (Participants) | 40 | 78
  Penis, Stage 3, Baseline | 0 | 1
  Penis, Stage 4, Baseline: number analyzed (Participants) | 40 | 78
  Penis, Stage 4, Baseline | 1 | 0
  Penis, Stage 5, Baseline: number analyzed (Participants) | 40 | 78
  Penis, Stage 5, Baseline | 0 | 0
  Penis, Stage 1, Week 17: number analyzed (Participants) | 40 | 77
  Penis, Stage 1, Week 17 | 29 | 68
  Penis, Stage 2, Week 17: number analyzed (Participants) | 40 | 77
  Penis, Stage 2, Week 17 | 10 | 8
  Penis, Stage 3, Week 17: number analyzed (Participants) | 40 | 77
  Penis, Stage 3, Week 17 | 0 | 1
  Penis, Stage 4, Week 17: number analyzed (Participants) | 40 | 77
  Penis, Stage 4, Week 17 | 1 | 0
  Penis, Stage 5, Week 17: number analyzed (Participants) | 40 | 77
  Penis, Stage 5, Week 17 | 0 | 0
  Penis, Stage 1, Week 33: number analyzed (Participants) | 36 | 75
  Penis, Stage 1, Week 33 | 22 | 58
  Penis, Stage 2, Week 33: number analyzed (Participants) | 36 | 75
  Penis, Stage 2, Week 33 | 11 | 16
  Penis, Stage 3, Week 33: number analyzed (Participants) | 36 | 75
  Penis, Stage 3, Week 33 | 3 | 1
  Penis, Stage 4, Week 33: number analyzed (Participants) | 36 | 75
  Penis, Stage 4, Week 33 | 0 | 0
  Penis, Stage 5, Week 33: number analyzed (Participants) | 36 | 75
  Penis, Stage 5, Week 33 | 0 | 0
  Penis, Stage 1, Week 49: number analyzed (Participants) | 37 | 72
  Penis, Stage 1, Week 49 | 21 | 57
  Penis, Stage 2, Week 49: number analyzed (Participants) | 37 | 72
  Penis, Stage 2, Week 49 | 9 | 14
  Penis, Stage 3, Week 49: number analyzed (Participants) | 37 | 72
  Penis, Stage 3, Week 49 | 5 | 1
  Penis, Stage 4, Week 49: number analyzed (Participants) | 37 | 72
  Penis, Stage 4, Week 49 | 2 | 0
  Penis, Stage 5, Week 49: number analyzed (Participants) | 37 | 72
  Penis, Stage 5, Week 49 | 0 | 0
  Testes, Stage 1, Baseline: number analyzed (Participants) | 40 | 78
  Testes, Stage 1, Baseline | 34 | 67
  Testes, Stage 2, Baseline: number analyzed (Participants) | 40 | 78
  Testes, Stage 2, Baseline | 4 | 10
  Testes, Stage 3, Baseline: number analyzed (Participants) | 40 | 78
  Testes, Stage 3, Baseline | 1 | 1
  Testes, Stage 4, Baseline: number analyzed (Participants) | 40 | 78
  Testes, Stage 4, Baseline | 1 | 0
  Testes, Stage 5, Baseline: number analyzed (Participants) | 40 | 78
  Testes, Stage 5, Baseline | 0 | 0
  Testes, Stage 1, Week 17: number analyzed (Participants) | 40 | 77
  Testes, Stage 1, Week 17 | 29 | 66
  Testes, Stage 2, Week 17: number analyzed (Participants) | 40 | 77
  Testes, Stage 2, Week 17 | 10 | 10
  Testes, Stage 3, Week 17: number analyzed (Participants) | 40 | 77
  Testes, Stage 3, Week 17 | 0 | 1
  Testes, Stage 4, Week 17: number analyzed (Participants) | 40 | 77
  Testes, Stage 4, Week 17 | 1 | 0
  Testes, Stage 5, Week 17: number analyzed (Participants) | 40 | 77
  Testes, Stage 5, Week 17 | 0 | 0
  Testes, Stage 1, Week 33: number analyzed (Participants) | 36 | 75
  Testes, Stage 1, Week 33 | 24 | 59
  Testes, Stage 2, Week 33: number analyzed (Participants) | 36 | 75
  Testes, Stage 2, Week 33 | 9 | 15
  Testes, Stage 3, Week 33: number analyzed (Participants) | 36 | 75
  Testes, Stage 3, Week 33 | 1 | 1
  Testes, Stage 4, Week 33: number analyzed (Participants) | 36 | 75
  Testes, Stage 4, Week 33 | 2 | 0
  Testes, Stage 5, Week 33: number analyzed (Participants) | 36 | 75
  Testes, Stage 5, Week 33 | 0 | 0
  Testes, Stage 1, Week 49: number analyzed (Participants) | 37 | 71
  Testes, Stage 1, Week 49 | 19 | 53
  Testes, Stage 2, Week 49: number analyzed (Participants) | 37 | 71
  Testes, Stage 2, Week 49 | 11 | 15
  Testes, Stage 3, Week 49: number analyzed (Participants) | 37 | 71
  Testes, Stage 3, Week 49 | 4 | 3
  Testes, Stage 4, Week 49: number analyzed (Participants) | 37 | 71
  Testes, Stage 4, Week 49 | 3 | 0
  Testes, Stage 5, Week 49: number analyzed (Participants) | 37 | 71
  Testes, Stage 5, Week 49 | 0 | 0

16. Primary Outcome: Number of Participants With Vital Signs Findings Reported as SAEs by Week 49
Description: Vital signs evaluation included supine systolic and diastolic blood pressure (BP), pulse rate, and respiratory rate. An SAE was any untoward medical occurrence at any dose that resulted in death; was life threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in congenital anomaly/birth defect. Investigators determined which vital signs findings were reported as SAEs.
Time Frame: Baseline to Week 49 visit
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Domagrozumab
Number analyzed (Participants) | 40 | 80
Participants | 0 | 0

17. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Data Meeting Pre-specified Criteria by Week 49
Description: Number of participants with ECG data meeting the following criteria are presented: 1) corrected QT interval using Fridericia's formula (QTcF interval) <450msec; 2) QTcF interval >=450 and <480msec; 3) QTcF interval >=480 and <500msec; 4) QTcF interval>=500msec; 5) QTcF interval increase from baseline<30msec; 6) QTcF interval increase from baseline >=30 and <60msec; 7) QTcF interval increase from baseline >=60msec.
Time Frame: Baseline to Week 49 visit
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Domagrozumab 5 mg/kg | Domagrozumab 20 mg/kg | Domagrozumab 40 mg/kg
Number analyzed (Participants) | 40 | 70 | 67 | 69
Participants
  QTcF interval <450msec | 40 | 70 | 67 | 68
  QTcF interval>=450 and <480msec | 0 | 0 | 0 | 1
  QTcF interval >=480 and <500msec | 0 | 0 | 0 | 0
  QTcF interval>=500msec | 0 | 0 | 0 | 0
  QTcF interval increase <30msec | 40 | 66 | 65 | 63
  QTcF interval increase >=30 and <60msec | 0 | 4 | 2 | 6
  QTcF interval increase >=60msec | 0 | 0 | 0 | 0

18. Primary Outcome: Change From Baseline in Left Ventricular Ejection Fraction (LVEF) as Compared to Placebo by Week 49
Description: The LVEF was the ratio of blood ejected during systole to blood in the ventricle at the end of diastole. LVEF was measured by cardiac magnetic resonance image (MRI) or echocardiogram. The same method of cardiac imaging was used consistently within a single participant. Cardiac MRIs were read by a central imaging vendor and echocardiograms were read locally at each site. The LVEF values measured by cardiac MRI and echocardiogram are combined in the following presentation. The analysis of covariance (ANCOVA) model was used to analyze the change from baseline for domagrozumab compared to placebo on LVEF. The baseline result, age, use of angiotensin receptor blocker (ARB)/beta blocker/angiotensin converting enzyme (ACE) inhibitor and treatment were included as fixed effects in the model.
Time Frame: Baseline to Week 49 visit
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Ratio of blood
Arm/Group | Placebo | Domagrozumab
Number analyzed (Participants) | 35 | 72
Ratio of blood | -0.063 (0.8464) | -1.356 (0.5620)
Statistical Analysis 1: Comparison: Placebo vs Domagrozumab; Test type: Superiority; p = 0.2088, ANCOVA — The significance level is 0.05; Mean Difference (Net) = 1.293, 95% CI 2-sided [-0.7343 to 3.3200], Standard Error of Mean 1.0220 — Least square mean difference was calculated by placebo minus domagrozumab

19. Primary Outcome: Height-adjusted Z-score of Lumbar Spine Bone Mineral Density Over Time by Week 49
Description: Bone mineral density (BMD) was evaluated by Dual energy X-ray Absorptiometry (DXA). The height adjusted Z-score presented below is the number of standard deviations which compares the BMD of the participant to the average BMD matched for their age, sex and ethnicity. If the Z-score was -2 standard deviations or lower, the result was "below the expected range for age". If the Z-score was above -2 standard deviations, the result was "within the expected range for age".
Time Frame: Screening and Week 49
Population: This analysis population included all participants who received at least 1 dose of investigational drug. Number analyzed refers to number of participants evaluable for specified rows of timepoints.
Measure: Mean (Standard Deviation); unit: Standard deviations
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3
Number analyzed (Participants) | 41 | 39 | 40
Standard deviations
  Screening: number analyzed (Participants) | 41 | 37 | 37
  Screening | -0.545151 (1.2845570) | -0.622784 (1.0778788) | -0.572650 (1.0283031)
  Week 49: number analyzed (Participants) | 37 | 35 | 36
  Week 49 | -0.683750 (1.0673420) | -0.401631 (1.0758951) | -0.489513 (1.0057285)

20. Primary Outcome: Bone Age to Chronological Age Ratio by Week 49
Description: Bone age assessment was evaluated by the ratio of the bone age to the chronological age using the X rays of the hand and wrist. Ratio of bone age to chronological age was calculated by bone age/chronological age at scan date. Chronological age at scan date was calculated by (scan date-date of birth+1)/365.25.
Time Frame: Screening, Weeks 17, 33 and 49
Population: This analysis population included all participants who received at least 1 dose of investigational drug. Number of participants analyzed signifies number of participants who were evaluable for this outcome measure. Number analyzed refers to number of participants evaluable for specified rows of timepoints.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo | Domagrozumab
Number analyzed (Participants) | 40 | 80
Ratio
  Screening | 0.809 (0.1656) | 0.762 (0.1650)
  Week 17: number analyzed (Participants) | 40 | 76
  Week 17 | 0.805 (0.1567) | 0.749 (0.1654)
  Week 33: number analyzed (Participants) | 39 | 76
  Week 33 | 0.790 (0.1614) | 0.750 (0.1589)
  Week 49: number analyzed (Participants) | 32 | 68
  Week 49 | 0.770 (0.1604) | 0.761 (0.1778)

21. Primary Outcome: Number of Participants With Suicidal Ideation and Suicidal Behavior Reported as AEs by Week 49
Description: An AE was any untoward medical occurrence in a clinical investigation participant administered a product; the event did not need to have a causal relationship with the treatment. The Columbia Suicide Severity Rating Scale (C-SSRS) was performed to identify the risk of suicide ideation or behavior. AEs of suicide ideation or behavior were determined by the investigator.
Time Frame: Baseline to Week 49 visit
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Domagrozumab
Number analyzed (Participants) | 40 | 80
Participants
  Suicidal ideation | 0 | 0
  Suicidal behavior | 0 | 0

22. Primary Outcome: Change From Baseline on the 4 Stair Climb (4SC) as Compared to Placebo at Weeks 17, 33 and 49
Description: The 4SC quantified the time required for a participant to ascend 4 standard steps. Mixed effect model for repeated measures (MMRM) was used to analyze the change from baseline on 4SC for domagrozumab compared to placebo. The baseline result, treatment, time and treatment by time interaction were included as fixed effects in the model. Participants were included as a random effect and the model was fit with an unstructured covariance for the repeated measures.
Time Frame: Baseline, Weeks 17, 33 and 49
Population: This analysis population included all participants randomized and who had received at least 1 dose of randomized treatment. Number of participants analyzed signifies number of participants who were evaluable for this outcome measure. Number analyzed refers to number of participants evaluable for specified rows of timeponts.
Measure: Least Squares Mean (Standard Error); unit: Seconds
Arm/Group | Placebo | Domagrozumab
Number analyzed (Participants) | 40 | 80
Seconds
  Week 17: number analyzed (Participants) | 39 | 74
  Week 17 | 1.6896 (0.6776) | 1.6051 (0.4814)
  Week 33: number analyzed (Participants) | 33 | 70
  Week 33 | 3.6407 (1.5837) | 4.2244 (1.1209)
  Week 49: number analyzed (Participants) | 32 | 63
  Week 49 | 8.0122 (3.03) | 8.2835 (2.1507)
Statistical Analysis 1: Comparison: Placebo vs Domagrozumab; Week 17; Test type: Superiority; p = 0.9191, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.0845, 95% CI 2-sided [-1.7354 to 1.5663] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 2: Comparison: Placebo vs Domagrozumab; Week 33; Test type: Superiority; p = 0.7642, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 0.5837, 95% CI 2-sided [-3.2978 to 4.4652] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 3: Comparison: Placebo vs Domagrozumab; Week 49; Test type: Superiority; p = 0.9423, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 0.2712, 95% CI 2-sided [-7.3799 to 7.9223] — Mean difference was calculated by domagrozumab minus placebo

23. Secondary Outcome: Change From Baseline as Compared to Placebo on Forced Vital Capacity (FVC) at Weeks 17, 33 and 49
Description: FVC was measured by spirometry to evaluate respiratory muscle function. MMRM was used to analyze the change from baseline on FVC for domagrozumab compared to placebo. The stratification factor, baseline result, treatment, time and treatment by time interaction were included as fixed effects in the model. Participants were included as a random effect and the model was fit with an unstructured covariance for the repeated measures.
Time Frame: Baseline, Weeks 17, 33 and 49
Population: This analysis population included all participants randomized and who had received at least 1 dose of randomized treatment. Number of participants analyzed signifies number of participants who were evaluable for this outcome measure. Number analyzed refers to number of participants evaluable for specified rows of timepoints.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | Domagrozumab
Number analyzed (Participants) | 40 | 80
Liters
  Week 17: number analyzed (Participants) | 40 | 78
  Week 17 | 0.0578 (0.0327) | 0.0578 (0.0250)
  Week 33: number analyzed (Participants) | 37 | 76
  Week 33 | 0.1008 (0.0385) | 0.0749 (0.0286)
  Week 49: number analyzed (Participants) | 38 | 74
  Week 49 | 0.1513 (0.0367) | 0.1092 (0.0278)
Statistical Analysis 1: Comparison: Placebo vs Domagrozumab; Week 17; Test type: Superiority; p = 0.9993, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 0, 95% CI 2-sided [-0.0693 to 0.0693] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 2: Comparison: Placebo vs Domagrozumab; Week 33; Test type: Superiority; p = 0.5464, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.0259, 95% CI 2-sided [-0.1107 to 0.0589] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 3: Comparison: Placebo vs Domagrozumab; Week 49; Test type: Superiority; p = 0.3041, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.0420, 95% CI 2-sided [-0.1227 to 0.0386] — Mean difference was calculated by domagrozumab minus placebo

24. Secondary Outcome: Change From Baseline as Compared to Placebo on the Northstar Ambulatory Assessment (NSAA) at Weeks 17, 33 and 49
Description: The NSAA is a 17-item test that measured gross motor function. Each individual item received a score of 0-unable to perform independently, 1-able to perform with assistance, or 2-able to perform without assistance. A total score was achieved by summing all the individual items. The total score could range from 0 to 34 (fully-independent function). MMRM was used to analyze the change from baseline for domagrozumab compared to placebo. The stratification factor, baseline result, treatment, time and treatment by time interaction were included as fixed effects in the model. Participants were included as a random effect and the model was fit with an unstructured covariance for the repeated measures.
Time Frame: Baseline, Weeks 17, 33 and 49
Population: as for outcome 23
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Domagrozumab
Number analyzed (Participants) | 40 | 80
Units on a scale
  Week 17: number analyzed (Participants) | 38 | 77
  Week 17 | -1.9 (0.8) | -1.1 (0.6)
  Week 33: number analyzed (Participants) | 38 | 75
  Week 33 | -4.5 (0.8) | -2.0 (0.6)
  Week 49: number analyzed (Participants) | 37 | 73
  Week 49 | -5.2 (0.9) | -3.6 (0.7)
Statistical Analysis 1: Comparison: Placebo vs Domagrozumab; Week 17; Test type: Superiority; p = 0.3522, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 0.8, 95% CI 2-sided [-0.9 to 2.5] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 2: Comparison: Placebo vs Domagrozumab; Week 33; Test type: Superiority; p = 0.0061, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 2.5, 95% CI 2-sided [0.7 to 4.2] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 3: Comparison: Placebo vs Domagrozumab; Test type: Superiority — Week 49; p = 0.1268, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 1.6, 95% CI 2-sided [-0.5 to 3.8] — Mean difference was calculated by domagrozumab minus placebo

25. Secondary Outcome: Change From Baseline as Compared to Placebo on the Ankle Range of Motion (ROM) at Weeks 17, 33 and 49
Description: ROM was evaluated by using goniometry to evaluate the loss of motion in the ankles. MMRM was used to analyze the change from baseline on ROM for domagrozumab compared to placebo. The stratification factor, baseline result, treatment, time and treatment by time interaction were included as fixed effects in the model. Participants were included as a random effect and the model was fit with an unstructured covariance for the repeated measures.
Time Frame: Baseline, Weeks 17, 33 and 49
Population: This analysis population included all participants randomized and who had received at least 1 dose of randomized treatment. Number of participants analyzed signifies number of participants who were evaluable for this outcome measure. Number analyzed refers to number of participants evaluable for specified rows of categories.
Measure: Least Squares Mean (Standard Error); unit: Degrees of passive dorsiflexion
Arm/Group | Placebo | Domagrozumab
Number analyzed (Participants) | 40 | 80
Degrees of passive dorsiflexion
  Left ankle, Week 17: number analyzed (Participants) | 40 | 78
  Left ankle, Week 17 | -1.0 (1.2) | -1.4 (0.9)
  Left ankle, Week 33: number analyzed (Participants) | 37 | 76
  Left ankle, Week 33 | -1.9 (1.2) | -1.7 (0.9)
  Left ankle, Week 49: number analyzed (Participants) | 38 | 75
  Left ankle, Week 49 | -2.3 (1.3) | -3.7 (1.0)
  Right ankle, Week 17: number analyzed (Participants) | 40 | 78
  Right ankle, Week 17 | -2.1 (1.3) | -1.3 (1.0)
  Right ankle, Week 33: number analyzed (Participants) | 37 | 76
  Right ankle, Week 33 | -4.1 (1.3) | -1.3 (0.9)
  Right ankle, Week 49: number analyzed (Participants) | 38 | 75
  Right ankle, Week 49 | -3.6 (1.4) | -3.6 (1.1)
Statistical Analysis 1: Comparison: Placebo vs Domagrozumab; Left ankle, Week 17; Test type: Superiority; p = 0.7337, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.4, 95% CI 2-sided [-2.9 to 2.1] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 2: Comparison: Placebo vs Domagrozumab; Left ankle, Week 33; Test type: Superiority; p = 0.8893, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 0.2, 95% CI 2-sided [-2.4 to 2.7] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 3: Comparison: Placebo vs Domagrozumab; Left ankle, Week 49; Test type: Superiority; p = 0.2939, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -1.5, 95% CI 2-sided [-4.3 to 1.3] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 4: Comparison: Placebo vs Domagrozumab; Right ankle, Week 17; Test type: Superiority; p = 0.5995, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 0.8, 95% CI 2-sided [-2.1 to 3.6] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 5: Comparison: Placebo vs Domagrozumab; Right ankle, Week 33; Test type: Superiority; p = 0.0385, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 2.9, 95% CI 2-sided [0.2 to 5.6] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 6: Comparison: Placebo vs Domagrozumab; Right ankle, Week 49; Test type: Superiority; p = 0.9927, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 0, 95% CI 2-sided [-3.3 to 3.2] — Mean difference was calculated by domagrozumab minus placebo

26. Secondary Outcome: Change From Baseline as Compared to Placebo on the Performance of Upper Limb (PUL) Overall Score at Weeks 17, 33 and 49
Description: The PUL was used to assess motor performance of the upper limb. The PUL scale includes 22 items; an entry item defining the starting functional level, and 21 items subdivided into three levels: shoulder (4 items), middle (9 items) and distal (8 items). Scoring options per item may not be uniform and may vary from 0-1 and 0-6, according to the performance, with higher values corresponding to better performance. A total maximum score of 74 is achieved by adding the individual level scores. MMRM was used to analyze the change from baseline for domagrozumab compared to placebo. The stratification factor, baseline result, treatment, time and treatment by time interaction were included as fixed effects in the model. Participants were included as a random effect and the model was fit with an unstructured covariance for the repeated measures.
Time Frame: Baseline, Weeks 17, 33 and 49
Population: as for outcome 23
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Domagrozumab
Number analyzed (Participants) | 40 | 80
Units on a scale
  Week 17: number analyzed (Participants) | 39 | 78
  Week 17 | -0.7 (0.6) | -1.0 (0.4)
  Week 33: number analyzed (Participants) | 37 | 76
  Week 33 | -2.7 (1.1) | -0.9 (0.8)
  Week 49: number analyzed (Participants) | 38 | 74
  Week 49 | -1.3 (0.5) | -1.4 (0.4)
Statistical Analysis 1: Comparison: Placebo vs Domagrozumab; Week 17; Test type: Superiority; p = 0.6049, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.3, 95% CI 2-sided [-1.7 to 1.0] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 2: Comparison: Placebo vs Domagrozumab; Week 33; Test type: Superiority; p = 0.2065, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 1.7, 95% CI 2-sided [-1.0 to 4.4] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 3: Comparison: Placebo vs Domagrozumab; Week 49; Test type: Superiority; p = 0.9391, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 0, 95% CI 2-sided [-1.3 to 1.2] — Mean difference was calculated by domagrozumab minus placebo

27. Secondary Outcome: Change From Baseline as Compared to Placebo on the Six Minute Walk Distance (6MWD) Score at Weeks 17, 33 and 49
Description: 6MWD evaluated ambulation ability by measuring the distance walked in 6 minutes. MMRM was used to analyze the change from baseline on 6MWD for domagrozumab compared to placebo. The stratification factor, baseline result, treatment, time and treatment by time interaction were included as fixed effects in the model. Participants were included as a random effect and the model was fit with an unstructured covariance for the repeated measures.
Time Frame: Baseline, Weeks 17, 33 and 49
Population: as for outcome 23
Measure: Least Squares Mean (Standard Error); unit: Meters
Arm/Group | Placebo | Domagrozumab
Number analyzed (Participants) | 40 | 80
Meters
  Week 17: number analyzed (Participants) | 36 | 74
  Week 17 | -32.0 (9.1) | -30.2 (6.9)
  Week 33: number analyzed (Participants) | 31 | 70
  Week 33 | -52.3 (9.9) | -43.4 (7.4)
  Week 49: number analyzed (Participants) | 30 | 61
  Week 49 | -56.5 (12.7) | -58.0 (9.3)
Statistical Analysis 1: Comparison: Placebo vs Domagrozumab; Week 17; Test type: Superiority; p = 0.8499, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 1.8, 95% CI 2-sided [-16.7 to 20.3] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 2: Comparison: Placebo vs Domagrozumab; Week 33; Test type: Superiority; p = 0.4008, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 8.9, 95% CI 2-sided [-12.0 to 29.8] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 3: Comparison: Placebo vs Domagrozumab; Week 49; Test type: Superiority; p = 0.9160, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -1.5, 95% CI 2-sided [-30.0 to 27.0] — Mean difference was calculated by domagrozumab minus placebo

28. Secondary Outcome: Change From Baseline as Compared to Placebo on Muscle Strength of Elbow Extension at Weeks 17, 33 and 49
Description: Muscle strength was quantified by means of a handheld dynamometer. The following muscle groups were evaluated: knee extension, elbow flexion, hip abduction, elbow extension and shoulder abduction. MMRM was used to analyze the change from baseline on muscle strength for domagrozumab compared to placebo. The stratification factor, baseline result, treatment, time and treatment by time interaction were included as fixed effects in the model. Participants were included as a random effect and the model was fit with an unstructured covariance for the repeated measures.
Time Frame: Baseline, Weeks 17, 33 and 49
Population: as for outcome 25
Measure: Least Squares Mean (Standard Error); unit: Kilograms
Arm/Group | Placebo | Domagrozumab
Number analyzed (Participants) | 40 | 80
Kilograms
  Left elbow extension, Week 17: number analyzed (Participants) | 40 | 76
  Left elbow extension, Week 17 | -0.182 (0.183) | -0.067 (0.141)
  Left elbow extension, Week 33: number analyzed (Participants) | 35 | 76
  Left elbow extension, Week 33 | -0.213 (0.187) | -0.376 (0.141)
  Left elbow extension, Week 49: number analyzed (Participants) | 37 | 74
  Left elbow extension, Week 49 | -0.353 (0.200) | -0.479 (0.150)
  Right elbow extension, Week 17: number analyzed (Participants) | 40 | 77
  Right elbow extension, Week 17 | -0.064 (0.209) | -0.086 (0.158)
  Right elbow extension, Week 33: number analyzed (Participants) | 35 | 75
  Right elbow extension, Week 33 | -0.052 (0.197) | -0.491 (0.148)
  Right elbow extension, Week 49: number analyzed (Participants) | 37 | 74
  Right elbow extension, Week 49 | -0.396 (0.192) | -0.562 (0.145)
Statistical Analysis 1: Comparison: Placebo vs Domagrozumab; Left elbow extension, Week 17; Test type: Superiority; p = 0.5726, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 0.115, 95% CI 2-sided [-0.287 to 0.517] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 2: Comparison: Placebo vs Domagrozumab; Left elbow extension, Week 33; Test type: Superiority; p = 0.4334, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.163, 95% CI 2-sided [-0.574 to 0.248] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 3: Comparison: Placebo vs Domagrozumab; Left elbow extension, Week 49; Test type: Superiority; p = 0.5767, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.126, 95% CI 2-sided [-0.573 to 0.321] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 4: Comparison: Placebo vs Domagrozumab; Right elbow extension, Week 17; Test type: Superiority; p = 0.9274, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.022, 95% CI 2-sided [-0.489 to 0.446] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 5: Comparison: Placebo; Right elbow extension, Week 33; Test type: Superiority; p = 0.0469, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.439, 95% CI 2-sided [-0.872 to -0.006] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 6: Comparison: Placebo vs Domagrozumab; Right elbow extension, Week 49; Test type: Superiority; p = 0.4362, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.166, 95% CI 2-sided [-0.587 to 0.255] — Mean difference was calculated by domagrozumab minus placebo

29. Secondary Outcome: Change From Baseline as Compared to Placebo on Muscle Strength of Elbow Flexion at Weeks 17, 33 and 49
Description: as for outcome 28
Time Frame: Baseline, Weeks 17, 33 and 49
Population: as for outcome 25
Measure: Least Squares Mean (Standard Error); unit: Kilograms
Arm/Group | Placebo | Domagrozumab
Number analyzed (Participants) | 40 | 80
Kilograms
  Left elbow flexion, Week 17: number analyzed (Participants) | 40 | 76
  Left elbow flexion, Week 17 | -0.096 (0.237) | -0.252 (0.181)
  Left elbow flexion, Week 33: number analyzed (Participants) | 35 | 76
  Left elbow flexion, Week 33 | -0.194 (0.244) | -0.497 (0.183)
  Left elbow flexion, Week 49: number analyzed (Participants) | 37 | 74
  Left elbow flexion, Week 49 | -0.573 (0.205) | -0.734 (0.159)
  Right elbow flexion, Week 17: number analyzed (Participants) | 40 | 77
  Right elbow flexion, Week 17 | -0.035 (0.220) | -0.118 (0.168)
  Right elbow flexion, Week 33: number analyzed (Participants) | 35 | 75
  Right elbow flexion, Week 33 | -0.057 (0.234) | -0.418 (0.175)
  Right elbow flexion, Week 49: number analyzed (Participants) | 37 | 74
  Right elbow flexion, Week 49 | -0.495 (0.199) | -0.684 (0.152)
Statistical Analysis 1: Comparison: Placebo vs Domagrozumab; Left elbow flexion, Week 17; Test type: Superiority; p = 0.5557, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.156, 95% CI 2-sided [-0.679 to 0.367] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 2: Comparison: Placebo vs Domagrozumab; Left elbow flexion, Week 33; Test type: Superiority; p = 0.2669, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.303, 95% CI 2-sided [-0.841 to 0.235] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 3: Comparison: Placebo vs Domagrozumab; Left elbow flexion, Week 49; Test type: Superiority; p = 0.4665, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.161, 95% CI 2-sided [-0.598 to 0.276] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 4: Comparison: Placebo vs Domagrozumab; Right elbow flexion, Week 17; Test type: Superiority; p = 0.7335, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.083, 95% CI 2-sided [-0.564 to 0.399] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 5: Comparison: Placebo vs Domagrozumab; Right elbow flexion, Week 33; Test type: Superiority; p = 0.1695, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.361, 95% CI 2-sided [-0.877 to 0.156] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 6: Comparison: Placebo vs Domagrozumab; Right elbow flexion, Week 49; Test type: Superiority; p = 0.3783, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.189, 95% CI 2-sided [-0.612 to 0.234] — Mean difference was calculated by domagrozumab minus placebo

30. Secondary Outcome: Change From Baseline as Compared to Placebo on Muscle Strength of Hip Abduction at Weeks 17, 33 and 49
Description: as for outcome 28
Time Frame: Baseline, Weeks 17, 33 and 49
Population: as for outcome 25
Measure: Least Squares Mean (Standard Error); unit: Kilograms
Arm/Group | Placebo | Domagrozumab
Number analyzed (Participants) | 40 | 80
Kilograms
  Left hip abduction, Week 17: number analyzed (Participants) | 40 | 77
  Left hip abduction, Week 17 | 0.430 (0.321) | -0.156 (0.245)
  Left hip abduction, Week 33: number analyzed (Participants) | 35 | 76
  Left hip abduction, Week 33 | -0.217 (0.318) | -0.171 (0.236)
  Left hip abduction, Week 49: number analyzed (Participants) | 37 | 75
  Left hip abduction, Week 49 | -0.097 (0.334) | -0.475 (0.251)
  Right hip abduction, Week 17: number analyzed (Participants) | 40 | 77
  Right hip abduction, Week 17 | 0.535 (0.320) | -0.154 (0.247)
  Right hip abduction, Week 33: number analyzed (Participants) | 35 | 76
  Right hip abduction, Week 33 | 0.087 (0.340) | -0.249 (0.255)
  Right hip abduction, Week 49: number analyzed (Participants) | 37 | 75
  Right hip abduction, Week 49 | 0.056 (0.343) | -0.266 (0.260)
Statistical Analysis 1: Comparison: Placebo vs Domagrozumab; Left hip abduction, Week 17; Test type: Superiority; p = 0.1078, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.586, 95% CI 2-sided [-1.303 to 0.130] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 2: Comparison: Placebo vs Domagrozumab; Left hip abduction, Week 33; Test type: Superiority; p = 0.8967, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 0.046, 95% CI 2-sided [-0.654 to 0.746] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 3: Comparison: Placebo vs Domagrozumab; Left hip abduction, Week 49; Test type: Superiority; p = 0.3196, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.378, 95% CI 2-sided [-1.128 to 0.371] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 4: Comparison: Placebo vs Domagrozumab; Right hip abduction, Week 17; Test type: Superiority; p = 0.0526, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.689, 95% CI 2-sided [-1.386 to 0.008] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 5: Comparison: Placebo vs Domagrozumab; Right hip abduction, Week 33; Test type: Superiority; p = 0.3739, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.336, 95% CI 2-sided [-1.082 to 0.410] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 6: Comparison: Placebo vs Domagrozumab; Right hip abduction, Week 49; Test type: Superiority; p = 0.4019, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.322, 95% CI 2-sided [-1.079 to 0.436] — Mean difference was calculated by domagrozumab minus placebo

31. Secondary Outcome: Change From Baseline as Compared to Placebo on Muscle Strength of Knee Extension at Weeks 17, 33 and 49
Description: as for outcome 28
Time Frame: Baseline, Weeks 17, 33 and 49
Population: as for outcome 25
Measure: Least Squares Mean (Standard Error); unit: Kilograms
Arm/Group | Placebo | Domagrozumab
Number analyzed (Participants) | 40 | 80
Kilograms
  Left knee extension, Week 17: number analyzed (Participants) | 40 | 77
  Left knee extension, Week 17 | -0.326 (0.336) | -0.434 (0.261)
  Left knee extension, Week 33: number analyzed (Participants) | 35 | 76
  Left knee extension, Week 33 | -0.713 (0.359) | -1.036 (0.272)
  Left knee extension, Week 49: number analyzed (Participants) | 37 | 75
  Left knee extension, Week 49 | -1.223 (0.369) | -1.110 (0.279)
  Right knee extension, Week 17: number analyzed (Participants) | 40 | 77
  Right knee extension, Week 17 | -0.213 (0.328) | -0.450 (0.253)
  Right knee extension, Week 33: number analyzed (Participants) | 35 | 76
  Right knee extension, Week 33 | -0.413 (0.380) | -0.880 (0.283)
  Right knee extension, Week 49: number analyzed (Participants) | 37 | 75
  Right knee extension, Week 49 | -0.976 (0.391) | -1.125 (0.292)
Statistical Analysis 1: Comparison: Placebo vs Domagrozumab; Left knee extension, Week 17; Test type: Superiority; p = 0.7676, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.107, 95% CI 2-sided [-0.825 to 0.610] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 2: Comparison: Placebo vs Domagrozumab; Left knee extension, Week 33; Test type: Superiority; p = 0.4127, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.322, 95% CI 2-sided [-1.098 to 0.454] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 3: Comparison: Placebo vs Domagrozumab; Left knee extension, Week 49; Test type: Superiority; p = 0.7815, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 0.113, 95% CI 2-sided [-0.693 to 0.919] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 4: Comparison: Placebo vs Domagrozumab; Right knee extension, Week 17; Test type: Superiority; p = 0.4975, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.236, 95% CI 2-sided [-0.924 to 0.451] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 5: Comparison: Placebo vs Domagrozumab; Right knee extension, Week 33; Test type: Superiority; p = 0.2646, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.467, 95% CI 2-sided [-1.294 to 0.359] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 6: Comparison: Placebo vs Domagrozumab; Right knee extension, Week 49; Test type: Superiority; p = 0.7320, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.149, 95% CI 2-sided [-1.008 to 0.710] — Mean difference was calculated by domagrozumab minus placebo

32. Secondary Outcome: Change From Baseline as Compared to Placebo on Muscle Strength of Shoulder Abduction at Weeks 17, 33 and 49
Description: as for outcome 28
Time Frame: Baseline, Weeks 17, 33 and 49
Population: as for outcome 25
Measure: Least Squares Mean (Standard Error); unit: Kilograms
Arm/Group | Placebo | Domagrozumab
Number analyzed (Participants) | 40 | 80
Kilograms
  Left shoulder abduction, Week 17: number analyzed (Participants) | 40 | 76
  Left shoulder abduction, Week 17 | -0.099 (0.213) | -0.143 (0.163)
  Left shoulder abduction, Week 33: number analyzed (Participants) | 35 | 76
  Left shoulder abduction, Week 33 | -0.123 (0.226) | -0.278 (0.166)
  Left shoulder abduction, Week 49: number analyzed (Participants) | 37 | 74
  Left shoulder abduction, Week 49 | -0.296 (0.238) | -0.319 (0.177)
  Right shoulder abduction, Week 17: number analyzed (Participants) | 39 | 77
  Right shoulder abduction, Week 17 | 0.079 (0.217) | -0.157 (0.165)
  Right shoulder abduction, Week 33: number analyzed (Participants) | 35 | 74
  Right shoulder abduction, Week 33 | 0.421 (0.251) | -0.336 (0.185)
  Right shoulder abduction, Week 49: number analyzed (Participants) | 37 | 74
  Right shoulder abduction, Week 49 | 0.140 (0.313) | -0.300 (0.229)
Statistical Analysis 1: Comparison: Placebo vs Domagrozumab; Left shoulder abduction, Week 17; Test type: Superiority; p = 0.8569, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.044, 95% CI 2-sided [-0.525 to 0.437] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 2: Comparison: Placebo vs Domagrozumab; Left shoulder abduction, Week 33; Test type: Superiority; p = 0.5495, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.154, 95% CI 2-sided [-0.663 to 0.355] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 3: Comparison: Placebo vs Domagrozumab; Left shoulder abduction, Week 49; Test type: Superiority; p = 0.9340, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.023, 95% CI 2-sided [-0.566 to 0.521] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 4: Comparison: Placebo vs Domagrozumab; Right shoulder abduction, Week 17; Test type: Superiority; p = 0.3279, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.236, 95% CI 2-sided [-0.711 to 0.239] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 5: Comparison: Placebo vs Domagrozumab; Right shoulder abduction, Week 33; Test type: Superiority; p = 0.0086, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.757, 95% CI 2-sided [-1.318 to -0.196] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 6: Comparison: Placebo vs Domagrozumab; Right shoulder abduction, Week 49; Test type: Superiority; p = 0.2328, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.439, 95% CI 2-sided [-1.165 to 0.286] — Mean difference was calculated by domagrozumab minus placebo

33. Secondary Outcome: Change From Baseline to Week 49 on 4SC for Participants in Sequence 3 Compared to the Natural History Control Group
Description: The 4SC quantified the time required for a participant to ascend 4 standard steps. MMRM was used to analyze the change from baseline on 4SC for the natural history control group compared to placebo group (Sequence 3). This MMRM was established to assess the appropriateness on using the natural history control group as a comparator. The natural history control group was established by filtering the CINRG (Cooperative International Neuromuscular Research Group) natural history database. Participants who met the following requirements at baseline and had evaluable 4SC data on Week 49 were included in this group: 1) age: 6 to <16 years; 2)treatment of glucocorticoid steroids >=6 months prior to baseline and continuous use until the latest visit week; 3) 4SC: 2-15.9 seconds; 4) participants who were ambulatory at baseline; 5) LVEF: >=55% or missing.
Time Frame: Baseline, Week 49
Population: This analysis population included all participants randomized in Sequence 3 and received at least 1 dose of randomized treatment. Number of participants analyzed signifies number of participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Seconds
Arm/Group | Sequence 3
Number analyzed (Participants) | 32
Seconds | 3.464 (1.232)
Statistical Analysis 1: Comparison: Sequence 3; Test type: Equivalence — The comparator was the natural history control group. The significance level is 0.05; p = 0.8908, Mixed Models Analysis; Mean Difference (Net) = 0.211, 95% CI 2-sided [-2.8353 to 3.2573] — Mean difference was calculated by Sequence 3 minus natural history control group

34. Secondary Outcome: Change From Baseline to Week 97 on 4SC for Participants in Sequence 1 Compared to the Natural History Control Group
Description: The 4SC quantified the time required for a participant to ascend 4 standard steps. MMRM was used to analyze the change from baseline on 4SC for domagrozumab compared to the natural history control group. The natural history control group was established by filtering the CINRG natural history database. Participants who met the following requirements at baseline and had evaluable 4SC data on Week 97 were included in this group: 1) age: 6 to <16 years; 2) treatment of glucocorticoid steroids >=6 months prior to baseline and continuous use until the latest visit week; 3) 4SC: 2-15.9 seconds; 4 participants who were ambulatory at baseline; 5) LVEF: >=55% or missing.
Time Frame: Baseline, Week 97
Population: This analysis population included all participants randomized in Sequence 1 and received at least 1 dose of randomized treatment. Number of participants analyzed signifies number of participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Seconds
Arm/Group | Sequence 1
Number analyzed (Participants) | 18
Seconds | 4.205 (1.011)
Statistical Analysis 1: Comparison: Sequence 1; Test type: Superiority — The comparator was the natural history control group. The significance level is 0.05; p = 0.4748, Mixed Models Analysis; Mean Difference (Net) = 0.819, 95% CI 2-sided [-1.4514 to 3.0895] — Mean difference was calculated by Sequence 1 minus natural history control group

35. Secondary Outcome: Change From Baseline to Week 49 on FVC for Participants in Sequence 3 Compared to the Natural History Control Group
Description: FVC was measured by spirometry to evaluate respiratory muscle function. MMRM was used to analyze the change from baseline on FVC for the natural history control group compared to placebo group (Sequence 3). MMRM was used to analyze the change from baseline on FVC for the natural history control group compared to placebo group (Sequence 3). This MMRM was established to assess the appropriateness on using the natural history control group as a comparator. The natural history control group was established by filtering the CINRG natural history database. Participants who met the following requirements at baseline and had evaluable FVC data on Week 49 were included in this group: 1) age: 6 to <16 years; 2)treatment of glucocorticoid steroids >=6 months prior to baseline and continuous use until the latest visit week; 3) 4SC: 2-15.9 seconds; 4) participants who were ambulatory at baseline; 5) LVEF: >=55% or missing.
Time Frame: Baseline, Week 49
Population: as for outcome 33
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Sequence 3
Number analyzed (Participants) | 38
Liters | 0.1358 (0.0328)
Statistical Analysis 1: Comparison: Sequence 3; Test type: Equivalence — The comparator was the natural history control group. The significance level is 0.05; p = 0.8070, Mixed Models Analysis; Mean Difference (Net) = 0.0097, 95% CI 2-sided [-0.0692 to 0.0887] — Mean difference was calculated by Sequence 3 minus natural history control group

36. Secondary Outcome: Change From Baseline to Week 97 on FVC for Participants in Sequence 1 Compared to the Natural History Control Group
Description: FVC was measured by spirometry to evaluate respiratory muscle function. MMRM was used to analyze the change from baseline on FVC for domagrozumab compared to the natural history control group. The natural history control group was established by filtering the CINRG natural history database. Participants who met the following requirements at baseline and had evaluable FVC data on Week 97 were included in this group: 1) age: 6 to <16 years; 2) treatment of glucocorticoid steroids >=6 months prior to baseline and continuous use until the latest visit week; 3) 4SC: 2-15.9 seconds; 4 participants who were ambulatory at baseline; 5) LVEF: >=55% or missing.
Time Frame: Baseline, Week 97
Population: as for outcome 34
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Sequence 1
Number analyzed (Participants) | 22
Liters | 0.2528 (0.0508)
Statistical Analysis 1: Comparison: Sequence 1; Test type: Superiority — The comparator was the natural history control group. The significance level is 0.05; p = 0.3643, Mixed Models Analysis; Mean Difference (Net) = 0.0506, 95% CI 2-sided [-0.0594 to 0.1607] — Mean difference was calculated by Sequence 1 minus natural history control group

37. Secondary Outcome: Change From Baseline to Week 49 on NSAA for Participants in Sequence 3 Compared to the Natural History Control Group
Description: The NSAA is a 17-item test that measured gross motor function. A total score could range from 0 to 34 (fully-independent function). MMRM was used to analyze the change from baseline on NSAA for the natural history control group compared to placebo group (Sequence 3). This MMRM was established to assess the appropriateness on the using natural history control group as a comparator. The natural history control group was established by filtering the CINRG natural history database. Participants who met the following requirements at baseline and had evaluable NSAA data on Week 49 were included in this group: 1) age: 6 to <16 years; 2)treatment of glucocorticoid steroids >=6 months prior to baseline and continuous use until the latest visit week; 3) 4SC: 2-15.9 seconds; 4) participants who were ambulatory at baseline; 5) LVEF: >=55% or missing.
Time Frame: Baseline, Week 49
Population: as for outcome 33
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Sequence 3
Number analyzed (Participants) | 37
Units on a scale | -4.8 (1.2)
Statistical Analysis 1: Comparison: Sequence 3; Test type: Equivalence — The comparator was the natural history control group. The significance level is 0.05; p = 0.0483, Mixed Models Analysis; Mean Difference (Net) = -2.9, 95% CI 2-sided [-5.7 to 0] — Mean difference was calculated by Sequence 3 minus natural history control group

38. Secondary Outcome: Change From Baseline to Week 97 on NSAA for Participants in Sequence 1 Compared to the Natural History Control Group
Description: The NSAA is a 17-item test that measured gross motor function. The total score could range from 0 to 34 (fully-independent function). MMRM was used to analyze the change from baseline on NSAA for domagrozumab compared to the natural history control group. The natural history control group was established by filtering the CINRG natural history database. Participants who met the following requirements at baseline and had evaluable NSAA data on Week 97 were included in this group: 1) age: 6 to <16 years; 2) treatment of glucocorticoid steroids >=6 months prior to baseline and continuous use until the latest visit week; 3) 4SC: 2-15.9 seconds; 4 participants who were ambulatory at baseline; 5) LVEF: >=55% or missing.
Time Frame: Baseline, Week 97
Population: as for outcome 34
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Sequence 1
Number analyzed (Participants) | 21
Units on a scale | -4.5 (1.2)
Statistical Analysis 1: Comparison: Sequence 1; Test type: Superiority — The comparator was the natural history control group. The significance level is 0.05; p = 0.0146, Mixed Models Analysis; Mean Difference (Net) = -3.9, 95% CI 2-sided [-7.0 to -0.8] — Mean difference was calculated by Sequence 1 minus natural history control group

39. Secondary Outcome: Change From Baseline to Week 49 on 6MWD for Participants in Sequence 3 Compared to the Natural History Control Group
Description: 6MWD evaluated ambulation ability by measuring the distance walked in 6 minutes. MMRM was used to analyze the change from baseline on 6MWD for the natural history control group compared to placebo group (Sequence 3). This MMRM was established to assess the appropriateness on using the natural history control group as a comparator. The natural history control group was established by filtering the CINRG natural history database. Participants who met the following requirements at baseline and had evaluable 6MWD data on Week 49 were included in this group: 1) age: 6 to <16 years; 2)treatment of glucocorticoid steroids >=6 months prior to baseline and continuous use until the latest visit week; 3) 4SC: 2-15.9 seconds; 4) participants who were ambulatory at baseline; 5) LVEF: >=55% or missing.
Time Frame: Baseline, Week 49
Population: as for outcome 33
Measure: Least Squares Mean (Standard Error); unit: Meters
Arm/Group | Sequence 3
Number analyzed (Participants) | 30
Meters | -80.8 (19.3)
Statistical Analysis 1: Comparison: Sequence 3; Test type: Equivalence — The comparator was the natural history control group. The significance level is 0.05; p = 0.1669, Mixed Models Analysis; Mean Difference (Net) = -31.6, 95% CI 2-sided [-76.9 to 13.6] — Mean difference was calculated by Sequence 3 minus natural history control group

40. Secondary Outcome: Change From Baseline to Week 97 on 6MWD for Participants in Sequence 1 Compared to the Natural History Control Group
Description: 6MWD evaluated ambulation ability by measuring the distance walked in 6 minutes. MMRM was used to analyze the change from baseline on 6MWD for domagrozumab compared to the natural history control group. The natural history control group was established by filtering the CINRG natural history database. Participants who met the following requirements at baseline and had evaluable 6MWD data on Week 97 were included in this group: 1) age: 6 to <16 years; 2)treatment of glucocorticoid steroids >=6 months prior to baseline and continuous use until the latest visit week; 3) 4SC: 2-15.9 seconds; 4) participants who were ambulatory at baseline; 5) LVEF: >=55% or missing.
Time Frame: Baseline, Week 97
Population: as for outcome 34
Measure: Least Squares Mean (Standard Error); unit: Meters
Arm/Group | Sequence 1
Number analyzed (Participants) | 17
Meters | -97.6 (20.7)
Statistical Analysis 1: Comparison: Sequence 1; Test type: Superiority — The comparator was the natural history control group. The significance level is 0.05; p = 0.0267, Mixed Models Analysis; Mean Difference (Net) = -66.3, 95% CI 2-sided [-124.5 to -8.1] — Mean difference was calculated by Sequence 1 minus natural history control group

41. Secondary Outcome: Change From Baseline as Compared to Placebo on 4SC at Week 17 in Pre-specified Subsets
Description: The 4SC quantified the time required for a participant to ascend 4 standard steps. A subset analysis was performed by categorizing participants into 3 subsets according to the baseline 4SC time: 1) <3.5 seconds, 2)>=3.5 seconds and <=8 seconds, 3) >8 seconds. MMRM was used to analyze the change from baseline for domagrozumab compared to placebo in subsets. The baseline result, treatment, time and treatment by time interaction were included as fixed effects in the model. Participants were included as a random effect and the model was fit with an unstructured covariance for the repeated measures.
Time Frame: Baseline, Week 17
Population: as for outcome 25
Measure: Least Squares Mean (Standard Error); unit: Seconds
Arm/Group | Placebo | Domagrozumab
Number analyzed (Participants) | 39 | 74
Seconds
  Baseline 4SC<3.5 seconds: number analyzed (Participants) | 11 | 28
  Baseline 4SC<3.5 seconds | 0.2329 (0.1513) | 0.1637 (0.092)
  Baseline 4SC>=3.5 and <=8 seconds: number analyzed (Participants) | 24 | 37
  Baseline 4SC>=3.5 and <=8 seconds | 0.7644 (0.4108) | 0.9758 (0.3283)
  Baseline 4SC>8 seconds: number analyzed (Participants) | 4 | 9
  Baseline 4SC>8 seconds | 7.7149 (4.8455) | 5.071 (3.0969)
Statistical Analysis 1: Comparison: Placebo vs Domagrozumab; Baseline 4SC<3.5 seconds; Test type: Superiority; p = 0.7033, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.0692, 95% CI 2-sided [-0.4345 to 0.2961] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 2: Comparison: Placebo vs Domagrozumab; Baseline 4SC>=3.5 and <= 8 seconds; Test type: Superiority; p = 0.6893, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 0.2114, 95% CI 2-sided [-0.8472 to 1.27] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 3: Comparison: Placebo vs Domagrozumab; Baseline 4SC>8 seconds; Test type: Superiority; p = 0.6469, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -2.6439, 95% CI 2-sided [-14.4292 to 9.1414] — Mean difference was calculated by domagrozumab minus placebo

42. Secondary Outcome: Change From Baseline as Compared to Placebo on 4SC at Week 33 in Pre-specified Subsets
Description: The 4SC quantified the time required for a participant to ascend 4 standard steps. A subset analysis was performed by categorizing participants into 3 subsets according to the baseline 4SC time: 1) <3.5 seconds, 2)>=3.5 seconds and <=8 seconds, 3) >8 seconds.MMRM was used to analyze the change from baseline for domagrozumab compared to placebo in subsets. The baseline result, treatment, time and treatment by time interaction were included as fixed effects in the model. Participants were included as a random effect and the model was fit with an unstructured covariance for the repeated measures.
Time Frame: Baseline, Week 33
Population: as for outcome 25
Measure: Least Squares Mean (Standard Error); unit: Seconds
Arm/Group | Placebo | Domagrozumab
Number analyzed (Participants) | 33 | 70
Seconds
  Baseline 4SC<3.5 seconds: number analyzed (Participants) | 9 | 29
  Baseline 4SC<3.5 seconds | 0.435 (0.1852) | 0.1062 (0.1061)
  Baseline 4SC>=3.5 and <=8 seconds: number analyzed (Participants) | 23 | 34
  Baseline 4SC>=3.5 and <=8 seconds | 2.2085 (0.8933) | 2.5542 (0.7234)
  Baseline 4SC>8 seconds: number analyzed (Participants) | 1 | 7
  Baseline 4SC>8 seconds | 3.7436 (8.1156) | 12.0329 (3.6174)
Statistical Analysis 1: Comparison: Placebo vs Domagrozumab; Baseline 4SC<3.5 seconds; Test type: Superiority; p = 0.1353, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.3289, 95% CI 2-sided [-0.7649 to 0.1072] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 2: Comparison: Placebo vs Domagrozumab; Baseline 4SC>=3.5 and <=8 seconds; Test type: Superiority; p = 0.7648, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 0.3457, 95% CI 2-sided [-1.9614 to 2.6528] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 3: Comparison: Placebo vs Domagrozumab; Baseline 4SC>8 seconds; Test type: Superiority; p = 0.3562, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 8.2893, 95% CI 2-sided [-9.6409 to 26.2194] — Mean difference was calculated by domagrozumab minus placebo

43. Secondary Outcome: Change From Baseline as Compared to Placebo on 4SC at Week 49 in Pre-specified Subsets
Description: as for outcome 41
Time Frame: Baseline, Week 49
Population: as for outcome 25
Measure: Least Squares Mean (Standard Error); unit: Seconds
Arm/Group | Placebo | Domagrozumab
Number analyzed (Participants) | 32 | 63
Seconds
  Baseline 4SC<3.5 seconds: number analyzed (Participants) | 11 | 28
  Baseline 4SC<3.5 seconds | 1.0056 (0.294) | 0.4474 (0.1816)
  Baseline 4SC>=3.5 and <= 8 seconds: number analyzed (Participants) | 20 | 30
  Baseline 4SC>=3.5 and <= 8 seconds | 3.526 (1.1574) | 3.6204 (0.9391)
  Baseline 4SC>8 seconds: number analyzed (Participants) | 1 | 5
  Baseline 4SC>8 seconds | 30.3411 (9.7373) | 19.053 (4.1965)
Statistical Analysis 1: Comparison: Placebo vs Domagrozumab; Baseline 4SC<3.5 seconds; Test type: Superiority; p = 0.1163, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.5582, 95% CI [-1.2615 to 0.1451] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 2: Comparison: Placebo vs Domagrozumab; Baseline 4SC>=3.5 and <=8 seconds; Test type: Superiority; p = 0.9503, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 0.0944, 95% CI 2-sided [-3.0798 to 3.2686] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 3: Comparison: Placebo vs Domagrozumab; Baseline 4SC>8 seconds; Test type: Superiority; p = 0.2947, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -11.2881, 95% CI 2-sided [-32.8328 to 10.2566] — Mean difference was calculated by domagrozumab minus placebo

44. Secondary Outcome: Change From Baseline as Compared to Placebo on FVC at Week 17 in Pre-specified Subsets
Description: FVC was measured by spirometry to evaluate respiratory muscle function. A subset analysis was performed by categorizing participants into 3 subsets according to the baseline 4SC time: 1) <3.5 seconds, 2)>=3.5 seconds and <=8 seconds, 3) >8 seconds. MMRM was used to analyze the change from baseline on FVC for domagrozumab compared to placebo in subsets. The stratification factor, baseline result, treatment, time and treatment by time interaction were included as fixed effects in the model. Participants were included as a random effect and the model was fit with an unstructured covariance for the repeated measures.
Time Frame: Baseline, Week 17
Population: as for outcome 25
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | Domagrozumab
Number analyzed (Participants) | 40 | 78
Liters
  Baseline 4SC<3.5 seconds: number analyzed (Participants) | 11 | 29
  Baseline 4SC<3.5 seconds | 0.0562 (0.0603) | 0.0722 (0.0368)
  Baseline 4SC>=3.5 and <=8 seconds: number analyzed (Participants) | 24 | 38
  Baseline 4SC>=3.5 and <=8 seconds | 0.0543 (0.0352) | 0.0411 (0.0276)
  Baseline 4SC>8 seconds: number analyzed (Participants) | 5 | 11
  Baseline 4SC>8 seconds | -0.0168 (0.0800) | 0.0721 (0.0534)
Statistical Analysis 1: Comparison: Placebo vs Domagrozumab; Baseline 4SC<3.5 seconds; Test type: Superiority; p = 0.8229, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 0.0159, 95% CI 2-sided [-0.1270 to 0.1588] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 2: Comparison: Placebo vs Domagrozumab; Baseline 4SC>=3.5 and <=8 seconds; Test type: Superiority; p = 0.7709, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.0132, 95% CI 2-sided [-0.1036 to 0.0772] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 3: Comparison: Placebo vs Domagrozumab; Baseline 4SC>8 seconds; Test type: Superiority; p = 0.3746, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 0.0889, 95% CI 2-sided [-0.1219 to 0.2996] — Mean difference was calculated by domagrozumab minus placebo

45. Secondary Outcome: Change From Baseline as Compared to Placebo on FVC at Week 33 in Pre-specified Subsets
Description: as for outcome 44
Time Frame: Baseline, Week 33
Population: as for outcome 25
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | Domagrozumab
Number analyzed (Participants) | 37 | 76
Liters
  Baseline 4SC<3.5 seconds: number analyzed (Participants) | 9 | 29
  Baseline 4SC<3.5 seconds | 0.1971 (0.0659) | 0.1036 (0.0389)
  Baseline 4SC>=3.5 and <=8 seconds: number analyzed (Participants) | 23 | 36
  Baseline 4SC>=3.5 and <=8 seconds | 0.0585 (0.0476) | 0.0468 (0.0376)
  Baseline 4SC>8 seconds: number analyzed (Participants) | 5 | 11
  Baseline 4SC>8 seconds | 0.0332 (0.1053) | 0.0895 (0.0703)
Statistical Analysis 1: Comparison: Placebo vs Domagrozumab; Baseline 4SC<3.5 seconds; Test type: Superiority; p = 0.2294, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.0934, 95% CI 2-sided [-0.2481 to 0.0613] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 2: Comparison: Placebo vs Domagrozumab; Baseline 4SC>=3.5 and <= 8 seconds; Test type: Superiority; p = 0.8485, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.0117, 95% CI 2-sided [-0.1339 to 0.1105] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 3: Comparison: Placebo vs Domagrozumab; Baseline 4SC>8 seconds; Test type: Superiority; p = 0.6645, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 0.0562, 95% CI 2-sided [-0.2187 to 0.3312] — Mean difference was calculated by domagrozumab minus placebo

46. Secondary Outcome: Change From Baseline as Compared to Placebo on FVC at Week 49 in Pre-specified Subsets
Description: as for outcome 44
Time Frame: Baseline, Week 49
Population: as for outcome 25
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | Domagrozumab
Number analyzed (Participants) | 38 | 74
Liters
  Baseline 4SC<3.5 seconds: number analyzed (Participants) | 11 | 28
  Baseline 4SC<3.5 seconds | 0.2199 (0.0675) | 0.1186 (0.0418)
  Baseline 4SC>=3.5 and <=8 seconds: number analyzed (Participants) | 22 | 35
  Baseline 4SC>=3.5 and <=8 seconds | 0.1364 (0.0376) | 0.1006 (0.0297)
  Baseline 4SC>8 seconds: number analyzed (Participants) | 5 | 11
  Baseline 4SC>8 seconds | 0.0052 (0.0936) | 0.1091 (0.0634)
Statistical Analysis 1: Comparison: Placebo vs Domagrozumab; Baseline 4SC<3.5 seconds; Test type: Superiority; p = 0.2101, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.1013, 95% CI 2-sided [-0.2622 to 0.0597] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 2: Comparison: Placebo vs Domagrozumab; Baseline 4SC>=3.5 and <= 8 seconds; Test type: Superiority; p = 0.4603, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.0359, 95% CI 2-sided [-0.1326 to 0.0608] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 3: Comparison: Placebo vs Domagrozumab; Baseline 4SC>8 seconds; Test type: Superiority; p = 0.3739, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 0.1039, 95% CI 2-sided [-0.1386 to 0.3463] — Mean difference was calculated by domagrozumab minus placebo

47. Secondary Outcome: Change From Baseline as Compared to Placebo on NSAA at Week 17 in Pre-specified Subsets
Description: The NSAA is a 17-item test that measured gross motor function. Each individual item received a score of 0-unable to perform independently, 1-able to perform with assistance, or 2-able to perform without assistance. A total score was achieved by summing all the individual items. The total score could range from 0 to 34 (fully-independent function). A subset analysis was performed by categorizing participants into 3 subsets according to the baseline 4SC time: 1) <3.5 seconds, 2)>=3.5 seconds and <=8 seconds, 3) >8 seconds. MMRM was used to analyze the change from baseline for domagrozumab compared to placebo in subsets. The stratification factor, baseline result, treatment, time and treatment by time interaction were included as fixed effects in the model. Participants were included as a random effect and the model was fit with an unstructured covariance for the repeated measures.
Time Frame: Baseline, Week 17
Population: as for outcome 25
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Domagrozumab
Number analyzed (Participants) | 38 | 77
Units on a scale
  Baseline 4SC<3.5 seconds: number analyzed (Participants) | 10 | 28
  Baseline 4SC<3.5 seconds | -0.4 (1.8) | -0.7 (1.1)
  Baseline 4SC>=3.5 and <=8 seconds: number analyzed (Participants) | 23 | 38
  Baseline 4SC>=3.5 and <=8 seconds | -1.3 (0.8) | -0.1 (0.6)
  Baseline 4SC>8 seconds: number analyzed (Participants) | 5 | 11
  Baseline 4SC>8 seconds | -3.2 (0.9) | -1.9 (0.6)
Statistical Analysis 1: Comparison: Placebo vs Domagrozumab; Baseline 4SC<3.5 seconds; Test type: Superiority; p = 0.8925, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.3, 95% CI 2-sided [-4.5 to 3.9] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 2: Comparison: Placebo vs Domagrozumab; Baseline 4SC>=3.5 and <=8 seconds; Test type: Superiority; p = 0.2107, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 1.2, 95% CI 2-sided [-0.7 to 3.2] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 3: Comparison: Placebo vs Domagrozumab; Baseline 4SC>8 seconds; Test type: Superiority; p = 0.2298, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 1.3, 95% CI 2-sided [-0.9 to 3.5] — Mean difference was calculated by domagrozumab minus placebo

48. Secondary Outcome: Change From Baseline as Compared to Placebo on NSAA at Week 33 in Pre-specified Subsets
Description: as for outcome 47
Time Frame: Baseline, Week 33
Population: as for outcome 25
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Domagrozumab
Number analyzed (Participants) | 38 | 75
Units on a scale
  Baseline 4SC<3.5 seconds: number analyzed (Participants) | 10 | 29
  Baseline 4SC<3.5 seconds | -3.9 (1.5) | -0.4 (0.9)
  Baseline 4SC>=3.5 and <=8 seconds: number analyzed (Participants) | 23 | 36
  Baseline 4SC>=3.5 and <=8 seconds | -3.5 (1.0) | -2.0 (0.8)
  Baseline 4SC>8 seconds: number analyzed (Participants) | 5 | 10
  Baseline 4SC>8 seconds | -5.6 (1.3) | -2.7 (0.9)
Statistical Analysis 1: Comparison: Placebo vs Domagrozumab; Baseline 4SC<3.5 seconds; Test type: Superiority; p = 0.0554, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 3.5, 95% CI 2-sided [-0.1 to 7.1] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 2: Comparison: Placebo vs Domagrozumab; Baseline 4SC>=3.5 and <= 8 seconds; Test type: Superiority; p = 0.2027, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 1.6, 95% CI 2-sided [-0.9 to 4.0] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 3: Comparison: Placebo vs Domagrozumab; Baseline 4SC>8 seconds; Test type: Superiority; p = 0.0926, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 2.9, 95% CI 2-sided [-0.5 to 6.3] — Mean difference was calculated by domagrozumab minus placebo

49. Secondary Outcome: Change From Baseline as Compared to Placebo on NSAA at Week 49 in Pre-specified Subsets
Description: as for outcome 47
Time Frame: Baseline, Week 49
Population: as for outcome 25
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Domagrozumab
Number analyzed (Participants) | 37 | 73
Units on a scale
  Baseline 4SC<3.5 seconds: number analyzed (Participants) | 11 | 29
  Baseline 4SC<3.5 seconds | -3.8 (1.8) | -1.8 (1.1)
  Baseline 4SC>=3.5 and <= 8 seconds: number analyzed (Participants) | 21 | 33
  Baseline 4SC>=3.5 and <= 8 seconds | -4.2 (1.1) | -3.7 (0.9)
  Baseline 4SC>8 seconds: number analyzed (Participants) | 5 | 11
  Baseline 4SC>8 seconds | -8.4 (1.4) | -4.4 (0.9)
Statistical Analysis 1: Comparison: Placebo vs Domagrozumab; Baseline 4SC<3.5 seconds; Test type: Superiority; p = 0.3597, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 2.0, 95% CI 2-sided [-2.4 to 6.3] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 2: Comparison: Placebo vs Domagrozumab; Baseline 4SC>=3.5 and <=8 seconds; Test type: Superiority; p = 0.7345, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 0.5, 95% CI 2-sided [-2.3 to 3.3] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 3: Comparison: Placebo vs Domagrozumab; Baseline 4SC>8 seconds; Test type: Superiority; p = 0.0320, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 4.0, 95% CI 2-sided [0.4 to 7.7] — Mean difference was calculated by domagrozumab minus placebo

50. Secondary Outcome: Change From Baseline as Compared to Placebo on PUL Overall Scores at Week 17 in Pre-specified Subsets
Description: The PUL was used to assess motor performance of the upper limb. The PUL scale includes 22 items; an entry item defining the starting functional level, and 21 items subdivided into three levels: shoulder (4 items), middle (9 items) and distal (8 items). Scoring options per item may not be uniform and may vary from 0-1 and 0-6, according to the performance, with higher values corresponding to better performance. A total maximum score of 74 is achieved by adding the individual level scores. A subset analysis was performed by categorizing participants into 3 subsets according to the baseline 4SC time. MMRM was used to analyze the change from baseline .The stratification factor, baseline result, treatment, time and treatment by time interaction were included as fixed effects in the model. Participants were included as a random effect and the model was fit with an unstructured covariance for the repeated measures.
Time Frame: Baseline, Week 17
Population: as for outcome 25
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Domagrozumab
Number analyzed (Participants) | 40 | 78
Units on a scale
  Baseline 4SC<3.5 seconds: number analyzed (Participants) | 11 | 29
  Baseline 4SC<3.5 seconds | -1.1 (1.1) | 0.2 (0.7)
  Baseline 4SC>=3.5 and <=8 seconds: number analyzed (Participants) | 23 | 38
  Baseline 4SC>=3.5 and <=8 seconds | 0.2 (0.7) | -1.0 (0.5)
  Baseline 4SC>8 seconds: number analyzed (Participants) | 5 | 11
  Baseline 4SC>8 seconds | 0.4 (1.7) | -0.5 (1.2)
Statistical Analysis 1: Comparison: Placebo vs Domagrozumab; Baseline 4SC<3.5 seconds; Test type: Superiority; p = 0.3345, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 1.2, 95% CI 2-sided [-1.3 to 3.8] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 2: Comparison: Placebo vs Domagrozumab; Baseline 4SC>=3.5 and <= 8 seconds; Test type: Superiority; p = 0.1400, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -1.2, 95% CI 2-sided [-2.9 to 0.4] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 3: Comparison: Placebo vs Domagrozumab; Baseline 4SC>8 seconds; Test type: Superiority; p = 0.6764, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.9, 95% CI 2-sided [-5.4 to 3.6] — Mean difference was calculated by domagrozumab minus placebo

51. Secondary Outcome: Change From Baseline as Compared to Placebo on PUL Overall Score at Week 33 in Pre-specified Subsets
Description: The PUL was used to assess motor performance of the upper limb. The PUL scale includes 22 items; an entry item defining the starting functional level, and 21 items subdivided into three levels: shoulder (4 items), middle (9 items) and distal (8 items).Scoring options per item may not be uniform and may vary from 0-1 and 0-6, according to the performance, with higher values corresponding to better performance. A total maximum score of 74 is achieved by adding the individual level scores. A subset analysis was performed by categorizing participants into 3 subsets according to the baseline 4SC time. MMRM was used to analyze the change from baseline.The stratification factor, baseline result, treatment, time and treatment by time interaction were included as fixed effects in the model. Participants were included as a random effect and the model was fit with an unstructured covariance for the repeated measures.
Time Frame: Baseline, Week 33
Population: as for outcome 25
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Domagrozumab
Number analyzed (Participants) | 37 | 76
Units on a scale
  Baseline 4SC<3.5 seconds: number analyzed (Participants) | 10 | 29
  Baseline 4SC<3.5 seconds | -6.4 (3.3) | 0.1 (2.0)
  Baseline 4SC>=3.5 and <= 8 seconds: number analyzed (Participants) | 22 | 36
  Baseline 4SC>=3.5 and <= 8 seconds | 0 (0.6) | -0.3 (0.5)
  Baseline 4SC>8 seconds: number analyzed (Participants) | 5 | 11
  Baseline 4SC>8 seconds | -1.0 (1.9) | -2.0 (1.2)
Statistical Analysis 1: Comparison: Placebo vs Domagrozumab; Baseline 4SC<3.5 seconds; Test type: Superiority; p = 0.0970, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 6.5, 95% CI 2-sided [-1.2 to 14.2] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 2: Comparison: Placebo vs Domagrozumab; Baseline 4SC>=3.5 and <=8 seconds; Test type: Superiority; p = 0.6919, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.3, 95% CI 2-sided [-1.9 to 1.3] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 3: Comparison: Placebo vs Domagrozumab; Baseline 4SC>8 seconds; Test type: Superiority; p = 0.6736, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -1.0, 95% CI 2-sided [-5.8 to 3.9] — Mean difference was calculated by domagrozumab minus placebo

52. Secondary Outcome: Change From Baseline as Compared to Placebo on PUL Overall Score at Week 49 in Pre-specified Subsets
Description: as for outcome 51
Time Frame: Baseline, Week 49
Population: as for outcome 25
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Domagrozumab
Number analyzed (Participants) | 38 | 75
Units on a scale
  Baseline 4SC<3.5 seconds: number analyzed (Participants) | 11 | 28
  Baseline 4SC<3.5 seconds | 0.3 (0.6) | 0.3 (0.4)
  Baseline 4SC>=3.5 and <=8 seconds: number analyzed (Participants) | 22 | 35
  Baseline 4SC>=3.5 and <=8 seconds | -0.9 (0.7) | -1.0 (0.5)
  Baseline 4SC>8 seconds: number analyzed (Participants) | 5 | 11
  Baseline 4SC>8 seconds | -2.6 (1.7) | -3.5 (1.1)
Statistical Analysis 1: Comparison: Placebo vs Domagrozumab; Baseline 4SC<3.5 seconds; Test type: Superiority; p = 0.9582, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 0, 95% CI 2-sided [-1.5 to 1.5] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 2: Comparison: Placebo vs Domagrozumab; Baseline 4SC>=3.5 and <= 8 seconds; Test type: Superiority; p = 0.8629, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.1, 95% CI 2-sided [-1.8 to 1.5] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 3: Comparison: Placebo vs Domagrozumab; Baseline 4SC>8 seconds; Test type: Superiority; p = 0.6746, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -0.9, 95% CI 2-sided [-5.5 to 3.7] — Mean difference was calculated by domagrozumab minus placebo

53. Secondary Outcome: Change From Baseline as Compared to Placebo on 6MWD at Week 17 in Pre-specified Subsets
Description: 6MWD evaluated ambulation ability by measuring the distance walked in 6 minutes. A subset analysis was performed by categorizing participants into 3 subsets according to the baseline 4SC time: 1) <3.5 seconds, 2)>=3.5 seconds and <=8 seconds, 3) >8 seconds. MMRM was used to analyze the change from baseline on 6MWD for domagrozumab compared to placebo in subsets. The stratification factor, baseline result, treatment, time and treatment by time interaction were included as fixed effects in the model. Participants were included as a random effect and the model was fit with an unstructured covariance for the repeated measures.
Time Frame: Baseline, Week 17
Population: as for outcome 25
Measure: Least Squares Mean (Standard Error); unit: Meters
Arm/Group | Placebo | Domagrozumab
Number analyzed (Participants) | 36 | 74
Meters
  Baseline 4SC<3.5 seconds: number analyzed (Participants) | 10 | 28
  Baseline 4SC<3.5 seconds | -6.9 (15.4) | -12.7 (9.3)
  Baseline 4SC>=3.5 and <=8 seconds: number analyzed (Participants) | 24 | 37
  Baseline 4SC>=3.5 and <=8 seconds | -21.0 (8.8) | -22.4 (7.0)
  Baseline 4SC>8 seconds: number analyzed (Participants) | 2 | 9
  Baseline 4SC>8 seconds | -34.0 (28.3) | -20.9 (16.3)
Statistical Analysis 1: Comparison: Placebo vs Domagrozumab; Baseline 4SC<3.5 seconds; Test type: Superiority; p = 0.7483, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -5.8, 95% CI 2-sided [-42.4 to 30.7] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 2: Comparison: Placebo vs Domagrozumab; Baseline 4SC>=3.5 and <=8 seconds; Test type: Superiority; p = 0.9053, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -1.3, 95% CI 2-sided [-23.9 to 21.2] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 3: Comparison: Placebo vs Domagrozumab; Baseline 4SC>8 seconds; Test type: Superiority; p = 0.6896, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 13.1, 95% CI 2-sided [-53.4 to 79.7] — Mean difference was calculated by domagrozumab minus placebo

54. Secondary Outcome: Change From Baseline as Compared to Placebo on 6MWD at Week 33 in Pre-specified Subsets
Description: as for outcome 53
Time Frame: Baseline, Week 33
Population: as for outcome 25
Measure: Least Squares Mean (Standard Error); unit: Meters
Arm/Group | Placebo | Domagrozumab
Number analyzed (Participants) | 31 | 70
Meters
  Baseline 4SC<3.5 seconds: number analyzed (Participants) | 9 | 29
  Baseline 4SC<3.5 seconds | -12.0 (13.2) | -15.7 (7.8)
  Baseline 4SC>=3.5 and <=8 seconds: number analyzed (Participants) | 21 | 34
  Baseline 4SC>=3.5 and <=8 seconds | -45.7 (10.9) | -38.4 (8.6)
  Baseline 4SC>8 seconds: number analyzed (Participants) | 1 | 7
  Baseline 4SC>8 seconds | -71.9 (40.6) | -55.6 (17.5)
Statistical Analysis 1: Comparison: Placebo vs Domagrozumab; Baseline 4SC<3.5 seconds; Test type: Superiority; p = 0.8117, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -3.7, 95% CI 2-sided [-34.8 to 27.5] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 2: Comparison: Placebo vs Domagrozumab; Baseline 4SC>=3.5 and <=8 seconds; Test type: Superiority; p = 0.6018, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 7.3, 95% CI 2-sided [-20.6 to 35.2] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 3: Comparison: Placebo vs Domagrozumab; Baseline 4SC>8 seconds; Test type: Superiority; p = 0.7152, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 16.3, 95% CI 2-sided [-73.4 to 106.0] — Mean difference was calculated by domagrozumab minus placebo

55. Secondary Outcome: Change From Baseline as Compared to Placebo on 6MWD at Week 49 in Pre-specified Subsets
Description: as for outcome 53
Time Frame: Baseline, Week 49
Population: as for outcome 25
Measure: Least Squares Mean (Standard Error); unit: Meters
Arm/Group | Placebo | Domagrozumab
Number analyzed (Participants) | 30 | 61
Meters
  Baseline 4SC<3.5 seconds: number analyzed (Participants) | 10 | 26
  Baseline 4SC<3.5 seconds | -33.5 (16.4) | -26.5 (10.1)
  Baseline 4SC>=3.5 and <=8 seconds: number analyzed (Participants) | 19 | 29
  Baseline 4SC>=3.5 and <=8 seconds | -42.0 (16.7) | -57.8 (13.4)
  Baseline 4SC>8 seconds: number analyzed (Participants) | 1 | 6
  Baseline 4SC>8 seconds | -75.1 (47.6) | -71.2 (18.9)
Statistical Analysis 1: Comparison: Placebo vs Domagrozumab; Baseline 4SC<3.5 seconds; Test type: Superiority; p = 0.7190, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 7.0, 95% CI 2-sided [-32.1 to 46.1] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 2: Comparison: Placebo vs Domagrozumab; Baseline 4SC>=3.5 and <=8 seconds; Test type: Superiority; p = 0.4634, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = -15.8, 95% CI 2-sided [-58.9 to 27.3] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 3: Comparison: Placebo vs Domagrozumab; Baseline 4SC>8 seconds; Test type: Superiority; p = 0.9400, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 3.9, 95% CI 2-sided [-100.7 to 108.5] — Mean difference was calculated by domagrozumab minus placebo

56. Secondary Outcome: Change From Baseline on Muscle Strength at Weeks 17, 33 and 49 in Pre-specified Subset (Baseline 4SC <3.5 Seconds)
Description: Muscle strength was quantified by means of a handheld dynamometer. The following muscle groups were evaluated: knee extension, elbow flexion, hip abduction, elbow extension and shoulder abduction. Change from baseline on muscle strength in all participants with baseline 4SC <3.5 seconds are presented below.
Time Frame: Baseline, Weeks 17, 33 and 49
Population: This analysis population included all participants (with baseline 4SC <3.5 seconds) randomized and who had received at least 1 dose o f randomized treatment. Number analyzed refers to number of participants evaluable for specified rows of categories.
Measure: Mean (95% Confidence Interval); unit: Kilograms
Arm/Group | Placebo | Domagrozumab
Number analyzed (Participants) | 11 | 30
Kilograms
  Left elbow extension, Week 17: number analyzed (Participants) | 11 | 27
  Left elbow extension, Week 17 | -0.08 [-0.811 to 0.647] | -0.33 [-0.960 to 0.301]
  Left elbow extension, Week 33: number analyzed (Participants) | 8 | 29
  Left elbow extension, Week 33 | -0.30 [-1.217 to 0.617] | -0.61 [-1.263 to 0.042]
  Left elbow extension, Week 49: number analyzed (Participants) | 10 | 28
  Left elbow extension, Week 49 | -1.13 [-2.130 to -0.130] | -0.60 [-1.304 to 0.097]
  Right elbow extension, Week 17: number analyzed (Participants) | 11 | 28
  Right elbow extension, Week 17 | 0.35 [-0.260 to 0.969] | -0.50 [-1.305 to 0.297]
  Right elbow extension, Week 33: number analyzed (Participants) | 8 | 29
  Right elbow extension, Week 33 | 0.46 [-0.681 to 1.606] | -0.88 [-1.591 to -0.168]
  Right elbow extension, Week 49: number analyzed (Participants) | 10 | 28
  Right elbow extension, Week 49 | -0.74 [-1.727 to 0.247] | -0.78 [-1.601 to 0.037]
  Left elbow flexion, Week 17: number analyzed (Participants) | 11 | 27
  Left elbow flexion, Week 17 | 0.65 [-0.290 to 1.600] | -0.61 [-1.602 to 0.387]
  Left elbow flexion, Week 33: number analyzed (Participants) | 8 | 29
  Left elbow flexion, Week 33 | 0.95 [-0.700 to 2.600] | -0.77 [-1.628 to 0.083]
  Left elbow flexion, Week 49: number analyzed (Participants) | 10 | 28
  Left elbow flexion, Week 49 | -0.88 [-1.664 to -0.096] | -0.96 [-1.857 to -0.057]
  Right elbow flexion, Week 17: number analyzed (Participants) | 11 | 28
  Right elbow flexion, Week 17 | 1.29 [0.401 to 2.181] | -0.21 [-0.938 to 0.517]
  Right elbow flexion, Week 33: number analyzed (Participants) | 8 | 29
  Right elbow flexion, Week 33 | 1.38 [-0.806 to 3.556] | -0.35 [-0.913 to 0.217]
  Right elbow flexion, Week 49: number analyzed (Participants) | 10 | 28
  Right elbow flexion, Week 49 | -0.33 [-1.082 to 0.422] | -0.69 [-1.310 to -0.061]
  Left hip abduction, Week 17: number analyzed (Participants) | 11 | 28
  Left hip abduction, Week 17 | 0.62 [-0.774 to 2.011] | -0.18 [-1.206 to 0.849]
  Left hip abduction, Week 33: number analyzed (Participants) | 8 | 29
  Left hip abduction, Week 33 | -0.51 [-2.235 to 1.210] | -0.02 [-0.835 to 0.786]
  Left hip abduction, Week 49: number analyzed (Participants) | 10 | 29
  Left hip abduction, Week 49 | -1.18 [-2.358 to -0.002] | -0.30 [-1.001 to 0.394]
  Right hip abduction, Week 17: number analyzed (Participants) | 11 | 28
  Right hip abduction, Week 17 | 1.47 [0.185 to 2.760] | -0.26 [-1.295 to 0.781]
  Right hip abduction, Week 33: number analyzed (Participants) | 8 | 29
  Right hip abduction, Week 33 | 0.40 [-0.739 to 1.539] | -0.34 [-1.172 to 0.496]
  Right hip abduction, Week 49: number analyzed (Participants) | 10 | 29
  Right hip abduction, Week 49 | -0.75 [-1.785 to 0.285] | -0.14 [-1.121 to 0.831]
  Left knee extension, Week 17: number analyzed (Participants) | 11 | 28
  Left knee extension, Week 17 | 0.99 [-0.192 to 2.174] | -1.12 [-2.186 to -0.050]
  Left knee extension, Week 33: number analyzed (Participants) | 8 | 29
  Left knee extension, Week 33 | 0.11 [-2.096 to 2.321] | -1.31 [-2.367 to -0.261]
  Left knee extension, Week 49: number analyzed (Participants) | 10 | 29
  Left knee extension, Week 49 | -1.54 [-3.308 to 0.228] | -1.33 [-2.516 to -0.140]
  Right knee extension, Week 17: number analyzed (Participants) | 11 | 28
  Right knee extension, Week 17 | 1.01 [-0.395 to 2.413] | -0.97 [-2.035 to 0.092]
  Right knee extension, Week 33: number analyzed (Participants) | 8 | 29
  Right knee extension, Week 33 | 0.26 [-1.037 to 1.562] | -1.31 [-2.494 to -0.120]
  Right knee extension, Week 49: number analyzed (Participants) | 10 | 29
  Right knee extension, Week 49 | -1.79 [-4.347 to 0.767] | -1.47 [-2.646 to -0.299]
  Left shoulder abduction, Week 17: number analyzed (Participants) | 11 | 27
  Left shoulder abduction, Week 17 | 0.66 [-0.218 to 1.545] | -0.33 [-0.866 to 0.206]
  Left shoulder abduction, Week 33: number analyzed (Participants) | 8 | 29
  Left shoulder abduction, Week 33 | 0.48 [-0.574 to 1.524] | -0.32 [-0.747 to 0.112]
  Left shoulder abduction, Week 49: number analyzed (Participants) | 10 | 28
  Left shoulder abduction, Week 49 | -0.32 [-1.357 to 0.717] | -0.16 [-0.627 to 0.306]
  Right shoulder abduction, Week 17: number analyzed (Participants) | 10 | 28
  Right shoulder abduction, Week 17 | 1.16 [0.421 to 1.899] | -0.40 [-1.058 to 0.258]
  Right shoulder abduction, Week 33: number analyzed (Participants) | 8 | 29
  Right shoulder abduction, Week 33 | 1.06 [-0.222 to 2.347] | -0.50 [-1.020 to 0.027]
  Right shoulder abduction, Week 49: number analyzed (Participants) | 10 | 28
  Right shoulder abduction, Week 49 | 0.17 [-0.749 to 1.089] | -0.20 [-0.852 to 0.445]

57. Secondary Outcome: Change From Baseline on Muscle Strength at Weeks 17, 33 and 49 in Pre-specified Subset (Baseline 4SC >=3.5 Seconds and <=8 Seconds)
Description: Muscle strength was quantified by means of a handheld dynamometer. The following muscle groups were evaluated: knee extension, elbow flexion, hip abduction, elbow extension and shoulder abduction. Change from baseline on muscle strength in all participants with baseline 4SC >=3.5 seconds and <=8 seconds are presented below.
Time Frame: Baseline, Weeks 17, 33 and 49
Population: This analysis population included all participants (with baseline 4SC >=3.5 seconds and <=8 seconds ) randomized and who had received at least 1 dose of randomized treatment. Number analyzed refers to number of participants evaluable for specified rows of categories.
Measure: Mean (95% Confidence Interval); unit: Kilograms
Arm/Group | Placebo | Domagrozumab
Number analyzed (Participants) | 24 | 38
Kilograms
  Left elbow extension, Week 17 | -0.05 [-0.353 to 0.244] | 0.31 [-0.073 to 0.689]
  Left elbow extension, Week 33: number analyzed (Participants) | 22 | 36
  Left elbow extension, Week 33 | -0.02 [-0.441 to 0.396] | -0.09 [-0.480 to 0.302]
  Left elbow extension, Week 49: number analyzed (Participants) | 22 | 35
  Left elbow extension, Week 49 | 0.15 [-0.223 to 0.532] | -0.26 [-0.803 to 0.289]
  Right elbow extension, Week 17 | 0 [-0.297 to 0.297] | 0.31 [-0.070 to 0.686]
  Right elbow extension, Week 33: number analyzed (Participants) | 22 | 35
  Right elbow extension, Week 33 | 0.02 [-0.367 to 0.412] | -0.17 [-0.558 to 0.209]
  Right elbow extension, Week 49: number analyzed (Participants) | 22 | 35
  Right elbow extension, Week 49 | -0.02 [-0.294 to 0.257] | -0.29 [-0.735 to 0.146]
  Left elbow flexion, Week 17 | -0.10 [-0.523 to 0.331] | 0.31 [-0.052 to 0.668]
  Left elbow flexion, Week 33: number analyzed (Participants) | 22 | 36
  Left elbow flexion, Week 33 | -0.26 [-0.598 to 0.071] | -0.13 [-0.515 to 0.254]
  Left elbow flexion, Week 49: number analyzed (Participants) | 22 | 35
  Left elbow flexion, Week 49 | -0.22 [-0.719 to 0.273] | -0.31 [-0.766 to 0.149]
  Right elbow flexion,Week 17 | -0.20 [-0.471 to 0.063] | 0.19 [-0.200 to 0.589]
  Right elbow flexion,Week 33: number analyzed (Participants) | 22 | 35
  Right elbow flexion,Week 33 | -0.15 [-0.529 to 0.239] | -0.23 [-0.682 to 0.225]
  Right elbow flexion,Week 49: number analyzed (Participants) | 22 | 35
  Right elbow flexion,Week 49 | -0.21 [-0.600 to 0.182] | -0.43 [-0.920 to 0.068]
  Left hip abduction, Week 17 | 0.65 [-0.019 to 1.319] | 0.34 [-0.134 to 0.823]
  Left hip abduction, Week 33: number analyzed (Participants) | 22 | 36
  Left hip abduction, Week 33 | -0.04 [-0.823 to 0.750] | -0.02 [-0.562 to 0.518]
  Left hip abduction, Week 49: number analyzed (Participants) | 22 | 35
  Left hip abduction, Week 49 | 0.48 [-0.336 to 1.290] | -0.09 [-1.042 to 0.865]
  Right hip abduction, Week 17 | 0.30 [-0.444 to 1.052] | 0.29 [-0.189 to 0.779]
  Right hip abduction, Week 33: number analyzed (Participants) | 22 | 36
  Right hip abduction, Week 33 | 0 [-1.062 to 1.071] | -0.05 [-0.655 to 0.555]
  Right hip abduction, Week 49: number analyzed (Participants) | 22 | 35
  Right hip abduction, Week 49 | 0.32 [-0.555 to 1.200] | 0.20 [-0.681 to 1.087]
  Left knee extension, Week 17 | -0.51 [-1.266 to 0.249] | 0.50 [-0.025 to 1.025]
  Left knee extension, Week 33: number analyzed (Participants) | 22 | 36
  Left knee extension, Week 33 | -0.59 [-1.576 to 0.404] | -0.67 [-1.339 to 0]
  Left knee extension, Week 49: number analyzed (Participants) | 22 | 35
  Left knee extension, Week 49 | -0.80 [-1.856 to 0.256] | -0.59 [-1.373 to 0.201]
  Right knee extension, Week 17 | -0.41 [-1.092 to 0.267] | 0.14 [-0.360 to 0.633]
  Right knee extension, Week 33: number analyzed (Participants) | 22 | 36
  Right knee extension, Week 33 | -0.35 [-1.227 to 0.536] | -0.53 [-1.237 to 0.170]
  Right knee extension, Week 49: number analyzed (Participants) | 22 | 35
  Right knee extension, Week 49 | -0.33 [-1.144 to 0.489] | -0.69 [-1.547 to 0.158]
  Left shoulder abduction, Week 17 | -0.24 [-0.757 to 0.274] | 0.49 [0.072 to 0.902]
  Left shoulder abduction, Week 33: number analyzed (Participants) | 22 | 36
  Left shoulder abduction, Week 33 | -0.19 [-0.552 to 0.170] | 0.03 [-0.442 to 0.503]
  Left shoulder abduction, Week 49: number analyzed (Participants) | 22 | 35
  Left shoulder abduction, Week 49 | -0.20 [-0.679 to 0.288] | -0.01 [-0.749 to 0.727]
  Rightshoulder abduction, Week 17 | -0.18 [-0.493 to 0.134] | 0.14 [-0.296 to 0.581]
  Right shoulder abduction, Week 33: number analyzed (Participants) | 22 | 34
  Right shoulder abduction, Week 33 | 0.38 [-0.260 to 1.014] | -0.18 [-0.683 to 0.319]
  Right shoulder abduction, Week 49: number analyzed (Participants) | 22 | 35
  Right shoulder abduction, Week 49 | 0.31 [-0.167 to 0.785] | -0.19 [-1.168 to 0.780]

58. Secondary Outcome: Change From Baseline on Muscle Strength at Weeks 17, 33 and 49 in Pre-specified Subset (Baseline 4SC >8 Seconds)
Description: Muscle strength was quantified by means of a handheld dynamometer. The following muscle groups were evaluated: knee extension, elbow flexion, hip abduction, elbow extension and shoulder abduction. Change from baseline on muscle strength in all participants with baseline 4SC >8 seconds are presented below.
Time Frame: Baseline, Weeks 17, 33 and 49
Population: This analysis population included all participants (with baseline 4SC >8 seconds) randomized and who had received at least 1 dose of randomized treatment. Number analyzed refers to number of participants evaluable for specified rows of categories.
Measure: Mean (95% Confidence Interval); unit: Kilograms
Arm/Group | Placebo | Domagrozumab
Number analyzed (Participants) | 5 | 12
Kilograms
  Left elbow extension, Week 17: number analyzed (Participants) | 5 | 11
  Left elbow extension, Week 17 | 0.10 [-0.665 to 0.865] | 0.14 [-0.226 to 0.498]
  Left elbow extension, Week 33: number analyzed (Participants) | 5 | 11
  Left elbow extension, Week 33 | 0.14 [-0.672 to 0.952] | 0.06 [-0.485 to 0.612]
  Left elbow extension, Week 49: number analyzed (Participants) | 5 | 11
  Left elbow extension, Week 49 | 0.08 [-0.380 to 0.540] | -0.15 [-0.456 to 0.146]
  Right elbow extension, Week 17: number analyzed (Participants) | 5 | 11
  Right elbow extension, Week 17 | 0.32 [-0.231 to 0.871] | 0.41 [0.099 to 0.719]
  Right elbow extension, Week 33: number analyzed (Participants) | 5 | 11
  Right elbow extension, Week 33 | 0.10 [-0.434 to 0.634] | 0.23 [-0.380 to 0.834]
  Right elbow extension, Week 49: number analyzed (Participants) | 5 | 11
  Right elbow extension, Week 49 | 0.06 [-0.275 to 0.395] | -0.13 [-0.467 to 0.213]
  Left elbow flexion, Week 17: number analyzed (Participants) | 5 | 11
  Left elbow flexion, Week 17 | -0.12 [-0.657 to 0.417] | 0.10 [-0.199 to 0.399]
  Left elbow flexion, Week 33: number analyzed (Participants) | 5 | 11
  Left elbow flexion, Week 33 | -0.36 [-1.108 to 0.388] | 0.33 [-0.684 to 1.339]
  Left elbow flexion, Week 49: number analyzed (Participants) | 5 | 11
  Left elbow flexion, Week 49 | -0.34 [-0.810 to 0.130] | -0.27 [-0.691 to 0.146]
  Right elbow flexion, Week 17: number analyzed (Participants) | 5 | 11
  Right elbow flexion, Week 17 | -0.30 [-0.933 to 0.333] | 0.20 [-0.168 to 0.568]
  Right elbow flexion, Week 33: number analyzed (Participants) | 5 | 11
  Right elbow flexion, Week 33 | -0.02 [-0.488 to 0.448] | 0.12 [-0.671 to 0.908]
  Right elbow flexion, Week 49: number analyzed (Participants) | 5 | 11
  Right elbow flexion, Week 49 | -0.14 [-0.567 to 0.287] | -0.34 [-0.646 to -0.027]
  Left hip abduction, Week 17: number analyzed (Participants) | 5 | 11
  Left hip abduction, Week 17 | 0.12 [-1.321 to 1.561] | -0.18 [-1.104 to 0.741]
  Left hip abduction, Week 33: number analyzed (Participants) | 5 | 11
  Left hip abduction, Week 33 | 0.36 [-1.232 to 1.952] | 0.65 [-1.112 to 2.403]
  Left hip abduction, Week 49: number analyzed (Participants) | 5 | 11
  Left hip abduction, Week 49 | 0.16 [-1.785 to 2.105] | -0.68 [-1.714 to 0.351]
  Right hip abduction, Week 17: number analyzed (Participants) | 5 | 11
  Right hip abduction, Week 17 | 0.22 [-0.698 to 1.138] | 0.09 [-0.546 to 0.728]
  Right hip abduction, Week 33: number analyzed (Participants) | 5 | 11
  Right hip abduction, Week 33 | 0.32 [-1.826 to 2.466] | 0.80 [-1.501 to 3.101]
  Right hip abduction, Week 49: number analyzed (Participants) | 5 | 11
  Right hip abduction, Week 49 | 0.68 [-1.743 to 3.103] | -0.55 [-1.569 to 0.460]
  Left knee extension, Week 17: number analyzed (Participants) | 5 | 11
  Left knee extension, Week 17 | 0.04 [-0.505 to 0.585] | 0.22 [-0.052 to 0.488]
  Left knee extension, Week 33: number analyzed (Participants) | 5 | 11
  Left knee extension, Week 33 | -0.24 [-1.188 to 0.708] | 0.32 [-0.749 to 1.386]
  Left knee extension, Week 49: number analyzed (Participants) | 5 | 11
  Left knee extension, Week 49 | -0.02 [-0.971 to 0.931] | -0.33 [-0.734 to 0.079]
  Right knee extension, Week 17: number analyzed (Participants) | 5 | 11
  Right knee extension, Week 17 | 0.32 [-0.442 to 1.082] | 0.17 [-0.204 to 0.549]
  Right knee extension, Week 33: number analyzed (Participants) | 5 | 11
  Right knee extension, Week 33 | -0.02 [-0.462 to 0.422] | 0.35 [-0.926 to 1.617]
  Right knee extension, Week 49: number analyzed (Participants) | 5 | 11
  Right knee extension, Week 49 | 0.06 [-0.410 to 0.530] | -0.20 [-0.564 to 0.164]
  Left shoulder abduction, Week 17: number analyzed (Participants) | 5 | 11
  Left shoulder abduction, Week 17 | 0.02 [-0.722 to 0.762] | -0.39 [-1.137 to 0.356]
  Left shoulder abduction, Week 33: number analyzed (Participants) | 5 | 11
  Left shoulder abduction, Week 33 | -0.12 [-0.692 to 0.452] | 0.29 [-1.461 to 2.042]
  Left shoulder abduction, Week 49: number analyzed (Participants) | 5 | 11
  Left shoulder abduction, Week 49 | 0.06 [-0.718 to 0.838] | -0.39 [-1.346 to 0.564]
  Right shoulder abduction, Week 17: number analyzed (Participants) | 5 | 11
  Right shoulder abduction, Week 17 | 0.14 [-0.820 to 1.100] | 0 [-0.568 to 0.568]
  Right shoulder abduction, Week 33: number analyzed (Participants) | 5 | 11
  Right shoulder abduction, Week 33 | 0.36 [-0.226 to 0.946] | 0.28 [-1.244 to 1.807]
  Right shoulder abduction, Week 49: number analyzed (Participants) | 5 | 11
  Right shoulder abduction, Week 49 | 0.32 [-0.357 to 0.997] | -0.17 [-1.132 to 0.787]

59. Secondary Outcome: Percent Change From Baseline in Whole Thigh Muscle Volume as Compared to Placebo by Weeks 17, 33 and 49
Description: The whole thigh muscle volume was measured by the proton density weighted sequence with magnetic resonance imaging (MRI) which was used to segment the entire thigh region into 3 primary regions for volumetric measure including 1) muscle; 2) inter/intra-muscular fat, 3) subcutaneous fat. MMRM was used to analyze the percent change from baseline for domagrozumab compared to placebo. The stratification factor, baseline result, treatment, time and treatment by time interaction were included as fixed effects in the model. Participants were included as a random effect and the model was fit with an unstructured covariance for the repeated measures.
Time Frame: Baseline, Weeks 17, 33 and 49
Population: This analysis population included all participants randomized and who had received at least 1 dose of randomized treatment. Number of participants analyzed signifies number of participants who were evaluable for this outcome measure. Number analyzed refers to number of participants evaluable for specified rows of time points.
Measure: Least Squares Mean (Standard Error); unit: Percent change of thigh muscle volume
Arm/Group | Placebo | Domagrozumab
Number analyzed (Participants) | 40 | 80
Percent change of thigh muscle volume
  Week 17: number analyzed (Participants) | 39 | 71
  Week 17 | 0.979 (1.062) | 3.924 (0.871)
  Week 33: number analyzed (Participants) | 37 | 70
  Week 33 | 1.380 (1.349) | 4.298 (1.043)
  Week 49: number analyzed (Participants) | 35 | 74
  Week 49 | -0.802 (1.623) | 3.285 (1.220)
Statistical Analysis 1: Comparison: Placebo vs Domagrozumab; Week 17; Test type: Superiority; p = 0.0087, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 2.945, 95% CI 2-sided [0.7597 to 5.1309] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 2: Comparison: Placebo vs Domagrozumab; Week 33; Test type: Superiority; p = 0.0536, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 2.918, 95% CI 2-sided [-0.0461 to 5.8811] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 3: Comparison: Placebo vs Domagrozumab; Week 49; Test type: Superiority; p = 0.0298, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 4.087, 95% CI 2-sided [0.4069 to 7.7677] — Mean difference was calculated by domagrozumab minus placebo

60. Secondary Outcome: Percent Change From Baseline as Compared to Placebo in Whole Thigh Muscle Volume Index by Weeks 17, 33 and 49
Description: The thigh muscle volume index was derived from the thigh muscle volume measurements as the fraction of total thigh tissue that was the lean muscle. MMRM was used to analyze the percent change from baseline for domagrozumab compared to placebo. The stratification factor, baseline result, treatment, time and treatment by time interaction were included as fixed effects in the model. Participants were included as a random effect and the model was fit with an unstructured covariance for the repeated measures.
Time Frame: Baseline, Weeks 17, 33 and 49
Population: as for outcome 25
Measure: Least Squares Mean (Standard Error); unit: Percent change of muscle volume index
Arm/Group | Placebo | Domagrozumab
Number analyzed (Participants) | 40 | 80
Percent change of muscle volume index
  Week 17: number analyzed (Participants) | 39 | 71
  Week 17 | -5.434 (0.844) | -3.859 (0.657)
  Week 33: number analyzed (Participants) | 37 | 70
  Week 33 | -9.408 (1.121) | -6.797 (0.836)
  Week 49: number analyzed (Participants) | 35 | 74
  Week 49 | -13.357 (1.358) | -10.149 (0.992)
Statistical Analysis 1: Comparison: Placebo vs Domagrozumab; Week 17; Test type: Superiority; p = 0.0684, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 1.575, 95% CI 2-sided [-0.1213 to 3.2715] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 2: Comparison: Placebo vs Domagrozumab; Week 33; Test type: Superiority; p = 0.0376, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 2.612, 95% CI 2-sided [0.1521 to 5.0711] — Mean difference was calculated by domagrozumab minus placebo
Statistical Analysis 3: Comparison: Placebo vs Domagrozumab; Week 49; Test type: Superiority; p = 0.0411, Mixed Models Analysis — The significance level is 0.05; Mean Difference (Net) = 3.208, 95% CI 2-sided [0.1318 to 6.2844] — Mean difference was calculated by domagrozumab minus placebo

61. Secondary Outcome: Change From Baseline in Whole Thigh Muscle Volume Through Week 97
Description: The whole thigh muscle volume was measured by the proton density weighted sequence with magnetic resonance imaging (MRI) which was used to segment the entire thigh region into 3 primary regions for volumetric measure including 1) muscle; 2) inter/intra-muscular fat, 3) subcutaneous fat.
Time Frame: Baseline, Weeks 17, 33, 49 and 97
Population: as for outcome 59
Measure: Mean (95% Confidence Interval); unit: Cubic centimeters
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3
Number analyzed (Participants) | 41 | 39 | 40
Cubic centimeters
  Muscle volume, Week 17: number analyzed (Participants) | 39 | 32 | 39
  Muscle volume, Week 17 | 36292.279 [14495.696 to 58088.862] | 26292.475 [5063.520 to 47521.430] | 5624.962 [-11939.656 to 23189.580]
  Muscle volume, Week 33: number analyzed (Participants) | 35 | 35 | 37
  Muscle volume, Week 33 | 37646.693 [8267.121 to 67026.264] | 37037.651 [10407.019 to 63668.283] | 12682.521 [-13221.920 to 38586.962]
  Muscle volume, Week 49: number analyzed (Participants) | 38 | 36 | 35
  Muscle volume, Week 49 | 37184.268 [1604.890 to 72763.647] | 25360.797 [-7334.654 to 58056.247] | -13438.274 [-45986.130 to 19109.581]
  Muscle volume, Week 97: number analyzed (Participants) | 21 | 22 | 18
  Muscle volume, Week 97 | 22715.921 [-47151.367 to 92583.210] | -42588.405 [-101774.836 to 16598.025] | -13903.138 [-85620.463 to 57814.187]

62. Secondary Outcome: Change From Baseline in Whole Thigh Muscle Volume Index Through Week 97
Description: The thigh muscle volume index was derived from the thigh muscle volume measurements as the fraction of total thigh tissue that was the lean muscle.
Time Frame: Baseline, Weeks 17, 33, 49 and 97
Population: as for outcome 59
Measure: Mean (95% Confidence Interval); unit: Percent of whole thign volume
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3
Number analyzed (Participants) | 41 | 39 | 40
Percent of whole thign volume
  Week 17: number analyzed (Participants) | 39 | 32 | 39
  Week 17 | -1.866 [-2.805 to -0.927] | -2.302 [-3.159 to -1.445] | -3.049 [-4.158 to -1.940]
  Week 33: number analyzed (Participants) | 35 | 35 | 37
  Week 33 | -4.151 [-5.629 to -2.672] | -3.706 [-5.016 to -2.396] | -5.582 [-7.016 to -4.149]
  Week 49: number analyzed (Participants) | 38 | 36 | 35
  Week 49 | -5.750 [-7.582 to -3.917] | -6.529 [-8.333 to -4.726] | -7.818 [-9.743 to -5.893]
  Week 97: number analyzed (Participants) | 21 | 22 | 18
  Week 97 | -12.130 [-16.597 to -7.662] | -14.861 [-19.379 to -10.344] | -14.906 [-19.042 to -10.769]

63. Secondary Outcome: Concentration of Growth Differentiation Factor 8 (GDF-8) at Time 0 (Pre-dose),(C0(GDF-8) )
Description: GDF-8, also called myostatin, is the target of domagrozumab. C0(GDF-8) was observed directly from data.
Time Frame: Predose on Day 1 of Week 1
Population: This analysis population included all enrolled participants in whom at least 1 GDF-8 concentration value was reported. Participants without contributing to the summary statistics are excluded below.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3
Number analyzed (Participants) | 40 | 39 | 39
Nanogram per milliliter (ng/mL) | 0.3187 (38773) | 0.4557 (6787) | 0.5052 (7405)

64. Secondary Outcome: Trough Serum Concentration of GDF-8 (Ctrough,(GDF-8)) for Participants Receiving Domagrozumab in Period 1
Description: GDF-8, also called myostatin, is the target of domagrozumab. Ctrough,(GDF-8) was observed directly from data.
Time Frame: Every 4 weeks on dosing day (at predose, end of 2-hour infusion and 6 hours since start of infusion) from Week 1 to Week 48
Population: This analysis population included all enrolled participants in Sequences 1 and 2 in whom at least 1 GDF-8 concentration value was reported. Participants without contributing to the summary statistics are excluded below.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Domagrozumab 5 mg/kg | Domagrozumab 20 mg/kg | Domagrozumab 40 mg/kg
Number analyzed (Participants) | 78 | 76 | 75
ng/mL | 4.540 (43) | 6.257 (42) | 7.449 (40)

65. Secondary Outcome: Ctrough,(GDF-8) for Participants of Sequence 3 in Period 2
Description: GDF-8, also called myostatin, is the target of domagrozumab. Ctrough,(GDF-8) was observed directly from data.
Time Frame: Every 4 weeks on dosing day (predose, end of 2-hour infusion and 6 hours since start of infusion) from Week 49 to Week 96
Population: This analysis population included all enrolled participants in Sequence 3 and in whom at least 1 GDF-8 concentration value was reported. Participants without contributing to the summary statistics are excluded below.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Domagrozumab 5 mg/kg: Participants received domagrozumab at a dose of 5 mg/kg over 2 hours by intravenous infusion every 4 weeks from Week 49 to Week 64 (4 doses).
- Domagrozumab 20 mg/kg: Participants received domagrozumab at a dose of 20 mg/kg over 2 hours by intravenous infusion every 4 weeks from Week 65 to Week 80 (4 doses).
- Domagrozumab 40 mg/kg: Participants received domagrozumab at a dose of 40 mg/kg over 2 hours by intravenous infusion every 4 weeks from Week 81 to Week 96 (4 doses).
Arm/Group | Domagrozumab 5 mg/kg | Domagrozumab 20 mg/kg | Domagrozumab 40 mg/kg
Number analyzed (Participants) | 37 | 30 | 21
ng/mL | 5.572 (36) | 7.776 (45) | 8.383 (53)

66. Secondary Outcome: Trough (Pre-dose) Serum Concentration (Ctrough) of Domagrozumab
Description: Ctrough was observed directly from data.
Time Frame: Every 4 weeks on dosing day (predose, end of 2-hour infusion and 6 hours since start of infusion) from Week 1 to Week 96 for Sequence 1; from Week 1 to Week 48 for Sequence 2; from Week 49 to Week 96 for Sequence 3
Population: This analysis population included all participants who received at least 1 dose of domagrozumab and in whom at least 1 concentration value was reported. Participants without contributing to the summary statistics are excluded below. Number analyzed refers to number of participants evaluable for specified rows of timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter (ug/mL)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3
Number analyzed (Participants) | 41 | 39 | 38
Microgram per milliliter (ug/mL)
  Week 1: number analyzed (Participants) | 0 | 1 | 0
  Week 1 |  | 75.3 (NA) — This is individual Ctrough value. Geometric coefficient of variation is not applicable. |
  Week 5: number analyzed (Participants) | 41 | 39 | 0
  Week 5 | 18.66 (28) | 19.26 (48) |
  Week 9: number analyzed (Participants) | 41 | 39 | 0
  Week 9 | 25.11 (32) | 27.95 (28) |
  Week 13: number analyzed (Participants) | 39 | 38 | 0
  Week 13 | 30.36 (28) | 31.98 (39) |
  Week 17: number analyzed (Participants) | 38 | 37 | 0
  Week 17 | 31.36 (30) | 35.08 (33) |
  Week 21: number analyzed (Participants) | 39 | 37 | 0
  Week 21 | 89.57 (43) | 97.5 (32) |
  Week 25: number analyzed (Participants) | 39 | 38 | 0
  Week 25 | 122.2 (25) | 129.4 (28) |
  Week 29: number analyzed (Participants) | 38 | 37 | 0
  Week 29 | 131.4 (26) | 140.4 (31) |
  Week 33: number analyzed (Participants) | 38 | 36 | 0
  Week 33 | 130.9 (36) | 148.2 (32) |
  Week 37: number analyzed (Participants) | 38 | 37 | 0
  Week 37 | 227.5 (33) | 250.7 (44) |
  Week 41: number analyzed (Participants) | 39 | 37 | 0
  Week 41 | 260.9 (31) | 284.5 (29) |
  Week 45: number analyzed (Participants) | 38 | 36 | 0
  Week 45 | 295.7 (32) | 323.4 (22) |
  Week 49: number analyzed (Participants) | 35 | 0 | 0
  Week 49 | 289.1 (31) |  |
  Week 53: number analyzed (Participants) | 37 | 0 | 38
  Week 53 | 307.3 (29) |  | 25.72 (36)
  Week 57: number analyzed (Participants) | 38 | 0 | 37
  Week 57 | 331.3 (29) |  | 39.9 (31)
  Week 61: number analyzed (Participants) | 38 | 0 | 36
  Week 61 | 327.6 (34) |  | 42.62 (46)
  Week 65: number analyzed (Participants) | 37 | 0 | 37
  Week 65 | 315.4 (39) |  | 48.39 (39)
  Week 69: number analyzed (Participants) | 34 | 0 | 34
  Week 69 | 315.7 (28) |  | 139.5 (47)
  Week 73: number analyzed (Participants) | 31 | 0 | 33
  Week 73 | 333.8 (34) |  | 168.1 (30)
  Week 77: number analyzed (Participants) | 30 | 0 | 30
  Week 77 | 309.6 (51) |  | 185.9 (27)
  Week 81: number analyzed (Participants) | 29 | 0 | 25
  Week 81 | 340.5 (26) |  | 201.2 (30)
  Week 85: number analyzed (Participants) | 25 | 0 | 25
  Week 85 | 367 (27) |  | 314.6 (32)
  Week 89: number analyzed (Participants) | 23 | 0 | 24
  Week 89 | 352.9 (26) |  | 367.4 (33)
  Week 93: number analyzed (Participants) | 22 | 0 | 20
  Week 93 | 380.2 (17) |  | 418.4 (33)

67. Secondary Outcome: Maximum Serum Concentration (Cmax) of Domagrozumab
Description: Cmax was observed directly from data.
Time Frame: as for outcome 66
Population: Data were not collected and analyzed due to study early termination.
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3
Number analyzed (Participants) | 0 | 0 | 0

68. Secondary Outcome: Time for Cmax (Tmax) of Domagrozumab
Description: Tmax was observed directly from the data.
Time Frame: as for outcome 66
Population: Data were not collected and analyzed due to study early termination.
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3
Number analyzed (Participants) | 0 | 0 | 0

69. Secondary Outcome: Terminal Half-life (t1/2) of Domagrozumab for Participants in Sequence 2 After the Last Dose of Domagrozumab
Description: t1/2 was calculated by Loge(2)/kel, where kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve. Participants in Sequence 2 received the last dose of domagrozumab at Week 45.
Time Frame: At predose, end of 2-hour infusion and 6 hours since start of infusion at Week 45
Population: Data were not collected and analyzed due to study early termination.
Arm/Group | Sequence 2
Number analyzed (Participants) | 0

70. Secondary Outcome: Area Under the Serum Concentration-time Curve Over the Dosing Interval Tau (AUCtau) of Domagrozumab
Description: The dosing interval tau was 672 hours (4 weeks). AUCtau was obtained by linear/log trapezoidal method. The AUCtau was assessed to fully characterize PK data and it was only assessed on the first 12 participants enrolled in the study who were required to complete additional PK visits.
Time Frame: At predose, end of 2-hour infusion,6 hours and 168 hours since start of infusion on Weeks 1, 13, 17, 29, 33 and 45
Population: This analysis population included participants who were among the first 12 participants enrolled in the study, had received at least 1 dose of domagrozumab and in whom at least 1 of the PK parameters of interest was calculated. Participants without contributing to the summary statistics are excluded below.
Measure: Median (Full Range); unit: Microgram*hour per milliliter (ug*hr/mL)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3
Number analyzed (Participants) | 2 | 5 | 0
Microgram*hour per milliliter (ug*hr/mL)
  Week 1 | 26500 [21700 to 31300] | 26300 [14700 to 31000] |
  Week 13 | 34650 [29500 to 39800] | 40500 [32300 to 50900] |
  Week 17: number analyzed (Participants) | 2 | 3 | 0
  Week 17 | 120500 [102000 to 139000] | 117000 [109000 to 128000] |
  Week 29: number analyzed (Participants) | 2 | 4 | 0
  Week 29 | 152000 [129000 to 175000] | 195500 [149000 to 197000] |
  Week 33: number analyzed (Participants) | 2 | 4 | 0
  Week 33 | 244500 [216000 to 273000] | 291000 [238000 to 372000] |
  Week 45: number analyzed (Participants) | 2 | 0 | 0
  Week 45 | 333500 [285000 to 382000] |  |

71. Secondary Outcome: Average Serum Concentration Over the Dosing Interval (Cav) of Domagrozumab
Description: Cav was calculated by AUCtau/tau. The Cav was assessed to fully characterize PK data and it was only assessed on the first 12 participants enrolled in the study who were required to complete additional PK visits.
Time Frame: At predose, end of 2-hour infusion, 6 hours and 168 hours since start of infusion on Weeks 1, 13, 17, 29, 33 and 45
Population: as for outcome 70
Measure: Median (Full Range); unit: ug/mL
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3
Number analyzed (Participants) | 2 | 5 | 0
ug/mL
  Week 1 | 39.45 [32.3 to 46.6] | 39.2 [21.9 to 46.1] |
  Week 13 | 51.55 [43.9 to 59.2] | 60.3 [48 to 75.7] |
  Week 17: number analyzed (Participants) | 2 | 3 | 0
  Week 17 | 179 [151 to 207] | 174 [162 to 191] |
  Week 29: number analyzed (Participants) | 2 | 4 | 0
  Week 29 | 226.5 [192 to 261] | 291 [221 to 293] |
  Week 33: number analyzed (Participants) | 2 | 4 | 0
  Week 33 | 364 [322 to 406] | 433.5 [354 to 553] |
  Week 45: number analyzed (Participants) | 2 | 0 | 0
  Week 45 | 496 [424 to 568] |  |

72. Secondary Outcome: Clearance (CL) of Domagrozumab
Description: CL was calculated by Dose/AUCtau. The CL was assessed to fully characterize PK data and it was only assessed on the first 12 participants enrolled in the study who were required to complete additional PK visits.
Time Frame: At predose, end of 2-hour infusion, 6 hours and 168 hours since start of infusion on Weeks 13, 29 and 45
Population: as for outcome 70
Measure: Median (Full Range); unit: Milliliter/hr/kilogram(mL/hr/kg)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3
Number analyzed (Participants) | 2 | 5 | 0
Milliliter/hr/kilogram(mL/hr/kg)
  Week 13 | 0.148 [0.126 to 0.17] | 0.123 [0.0983 to 0.155] |
  Week 29: number analyzed (Participants) | 2 | 4 | 0
  Week 29 | 0.1345 [0.114 to 0.155] | 0.102 [0.102 to 0.134] |
  Week 45: number analyzed (Participants) | 2 | 0 | 0
  Week 45 | 0.1225 [0.105 to 0.14] |  |

73. Secondary Outcome: Volume of Distribution at Steady State (Vss) of Domagrozumab for Participants in Sequence 2 Required for Additional PK Assessment
Description: Vss was calculated by CL*MRT, where MRT was the mean residence time. Vss was assessed to fully characterize PK data.
Time Frame: At predose, end of 2-hour infusion, 6 hours and 168 hours since start of infusion on Week 45
Population: Data were not collected and analyzed due to study early termination.
Arm/Group | Sequence 2
Number analyzed (Participants) | 0

74. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADA) Development by Week 97
Description: The criterion for positive result of ADA samples was ADA titer >=1.88.
Time Frame: Baseline, every 4 weeks from Week 5 to Week 97 visit or early termination
Population: This analysis population included all participants who received at least 1 dose of investigational drug. Number analyzed refers to the number of participants evaluable for specified rows of time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3
Number analyzed (Participants) | 41 | 39 | 40
Participants
  Baseline: number analyzed (Participants) | 40 | 39 | 0
  Baseline | 0 | 0 |
  Week 5: number analyzed (Participants) | 40 | 38 | 0
  Week 5 | 0 | 0 |
  Week 9: number analyzed (Participants) | 41 | 38 | 0
  Week 9 | 0 | 0 |
  Week 13: number analyzed (Participants) | 40 | 38 | 0
  Week 13 | 0 | 0 |
  Week 17: number analyzed (Participants) | 40 | 38 | 0
  Week 17 | 0 | 0 |
  Week 21: number analyzed (Participants) | 39 | 38 | 0
  Week 21 | 0 | 0 |
  Week 25: number analyzed (Participants) | 39 | 37 | 0
  Week 25 | 0 | 0 |
  Week 29: number analyzed (Participants) | 38 | 38 | 0
  Week 29 | 0 | 0 |
  Week 33: number analyzed (Participants) | 38 | 38 | 0
  Week 33 | 0 | 0 |
  Week 37: number analyzed (Participants) | 37 | 37 | 0
  Week 37 | 0 | 0 |
  Week 41: number analyzed (Participants) | 38 | 37 | 0
  Week 41 | 0 | 0 |
  Week 45: number analyzed (Participants) | 38 | 37 | 0
  Week 45 | 0 | 0 |
  Week 49: number analyzed (Participants) | 37 | 1 | 38
  Week 49 | 0 | 0 | 0
  Week 53: number analyzed (Participants) | 38 | 0 | 38
  Week 53 | 0 |  | 0
  Week 57: number analyzed (Participants) | 38 | 0 | 37
  Week 57 | 0 |  | 0
  Week 61: number analyzed (Participants) | 38 | 0 | 37
  Week 61 | 0 |  | 0
  Week 65: number analyzed (Participants) | 36 | 0 | 37
  Week 65 | 0 |  | 1
  Week 69: number analyzed (Participants) | 35 | 0 | 35
  Week 69 | 0 |  | 0
  Week 73: number analyzed (Participants) | 33 | 0 | 33
  Week 73 | 0 |  | 0
  Week 77: number analyzed (Participants) | 31 | 0 | 30
  Week 77 | 0 |  | 0
  Week 81: number analyzed (Participants) | 29 | 0 | 27
  Week 81 | 0 |  | 0
  Week 85: number analyzed (Participants) | 26 | 0 | 25
  Week 85 | 0 |  | 0
  Week 89: number analyzed (Participants) | 24 | 0 | 24
  Week 89 | 0 |  | 0
  Week 93: number analyzed (Participants) | 24 | 0 | 21
  Week 93 | 0 |  | 0
  Week 97: number analyzed (Participants) | 20 | 1 | 21
  Week 97 | 0 | 0 | 0
  Early termination: number analyzed (Participants) | 14 | 1 | 12
  Early termination | 0 | 0 | 0

75. Other Pre Specified Outcome: Area Under the Curve From Time Zero to Last Quantifiable Serum Concentration (AUClast) of Domagrozumab
Description: AUClast was calculated by linear/log trapezoidal method. AUCtau was obtained by linear/log trapezoidal method. AUClast was assessed to fully characterize PK data and it was only assessed on the first 12 participants enrolled in the study who were required to complete additional PK visits.
Time Frame: At predose, end of 2-hour infusion, 6 hours and 168 hours since start of infusion on Weeks 1, 13, 17, 29, 33 and 45
Population: Data were not collected and analyzed due to study early termination.
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 105 weeks
Description: The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs.
Groups:
- Domagrozumab 5 mg/kg, Period 1: Participants received domagrozumab at a dose of 5 mg/kg over 2 hours by intravenous infusion every 4 weeks from Week 1 to Week 16 (4 doses).
- Domagrozumab 20 mg/kg, Period 1: Participants received domagrozumab at a dose of 20 mg/kg over 2 hours by intravenous infusion every 4 weeks from Week 17 to Week 32 (4 doses).
- Domagrozumab 40 mg/kg, Period 1: Participants received domagrozumab at a dose of 40 mg/kg over 2 hours by intravenous infusion every 4 weeks from Week 33 to Week 48 (4 doses).
- Placebo, Period 1: Participants received placebo from Week 1 to Week 48.
- Domagrozumab 5 mg/kg, Period 2: Participants received domagrozumab at a dose of 5 mg/kg over 2 hours by intravenous infusion every 4 weeks from Week 49 to Week 64 (4 doses).
- Domagrozumab 20 mg/kg, Period 2: Participants received domagrozumab at a dose of 20 mg/kg over 2 hours by intravenous infusion every 4 weeks from Week 65 to Week 80 (4 doses).
- Domagrozumab 40 mg/kg, Period 2: Participants received domagrozumab at a dose of 40 mg/kg over 2 hours by intravenous infusion every 4 weeks from Week 81 to Week 96 (4 doses).
- Placebo, Period 2: Participants received placebo from Week 49 to Week 96.
Arm/Group | Domagrozumab 5 mg/kg, Period 1 | Domagrozumab 20 mg/kg, Period 1 | Domagrozumab 40 mg/kg, Period 1 | Placebo, Period 1 | Domagrozumab 5 mg/kg, Period 2 | Domagrozumab 20 mg/kg, Period 2 | Domagrozumab 40 mg/kg, Period 2 | Placebo, Period 2
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/78 | 0/76 | 0/40 | 0/38 | 0/38 | 0/66 | 0/37
Serious Adverse Events (participants affected / at risk) | 1/80 | 1/78 | 1/76 | 0/40 | 1/38 | 1/38 | 1/66 | 0/37
Other Adverse Events (participants affected / at risk) | 58/80 | 43/78 | 50/76 | 38/40 | 29/38 | 22/38 | 49/66 | 29/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Domagrozumab 5 mg/kg, Period 1 (N=80) | Domagrozumab 20 mg/kg, Period 1 (N=78) | Domagrozumab 40 mg/kg, Period 1 (N=76) | Placebo, Period 1 (N=40) | Domagrozumab 5 mg/kg, Period 2 (N=38) | Domagrozumab 20 mg/kg, Period 2 (N=38) | Domagrozumab 40 mg/kg, Period 2 (N=66) | Placebo, Period 2 (N=37)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Superior sagittal sinus thrombosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Domagrozumab 5 mg/kg, Period 1 (N=80) | Domagrozumab 20 mg/kg, Period 1 (N=78) | Domagrozumab 40 mg/kg, Period 1 (N=76) | Placebo, Period 1 (N=40) | Domagrozumab 5 mg/kg, Period 2 (N=38) | Domagrozumab 20 mg/kg, Period 2 (N=38) | Domagrozumab 40 mg/kg, Period 2 (N=66) | Placebo, Period 2 (N=37)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (8) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (6) | 3 (4) | 3 (4) | 4 (5) | 2 (2) | 2 (2) | 3 (6) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 4 (5) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (3) | 2 (2) | 7 (10) | 3 (4) | 0 (0) | 7 (9) | 5 (6)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 5 (5) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 8 (9) | 6 (7) | 6 (7) | 9 (13) | 3 (3) | 1 (1) | 4 (4) | 8 (13)
Chest pain (General disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (6) | 1 (2) | 1 (1) | 3 (5) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Gait inability (General disorders) | 2 (2) | 2 (2) | 1 (1) | 5 (5) | 1 (1) | 2 (2) | 3 (3) | 6 (6)
Infusion site swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 6 (9) | 6 (6) | 5 (5) | 9 (15) | 2 (2) | 1 (1) | 6 (8) | 2 (2)
Ear infection (Infections and infestations) | 3 (3) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 4 (4) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 3 (4) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (2) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 6 (6) | 3 (3)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 16 (18) | 13 (14) | 8 (10) | 11 (21) | 6 (6) | 3 (5) | 8 (11) | 9 (12)
Upper resiratory tract infection (Infections and infestations) | 6 (7) | 5 (5) | 7 (8) | 6 (13) | 5 (5) | 1 (1) | 9 (11) | 7 (7)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 3 (4) | 3 (4) | 1 (1) | 0 (0) | 3 (4) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 22 (32) | 15 (22) | 12 (13) | 20 (43) | 9 (18) | 7 (12) | 17 (28) | 7 (13)
Ligment sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 4 (4) | 4 (4)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 4 (4) | 3 (3) | 6 (10) | 4 (4) | 2 (2) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 4 (4) | 1 (1) | 6 (7) | 1 (2) | 0 (0) | 5 (5) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 11 (18) | 6 (9) | 6 (10) | 14 (24) | 4 (5) | 5 (7) | 11 (20) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (6) | 3 (3) | 3 (3) | 7 (9) | 5 (5) | 3 (3) | 4 (5) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1) | 4 (4) | 3 (3) | 3 (3) | 4 (4) | 10 (13) | 4 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (9) | 7 (14) | 3 (14) | 4 (5) | 2 (3) | 0 (0) | 3 (14) | 3 (13)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5) | 6 (6) | 6 (8) | 1 (1) | 0 (0) | 8 (10) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 3 (3) | 5 (6) | 1 (1) | 2 (2) | 4 (5) | 3 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (3) | 0 (0) | 6 (6) | 0 (0) | 1 (1) | 7 (9) | 3 (3)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 6 (6) | 0 (0) | 2 (2) | 5 (6) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was terminated because the primary efficacy objective (the efficacy of treatment with domagrozumab based on a mean change from baseline on 4 Stair Climb as compared to placebo following 48 weeks of treatment) was not met.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2016-08-15): https://cdn.clinicaltrials.gov/large-docs/63/NCT02310763/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-11): https://cdn.clinicaltrials.gov/large-docs/63/NCT02310763/SAP_001.pdf